Version Date: 05.12.2023

**Abbreviated Title:** Combo Immunotx in HPV Cancers

NIH Protocol #: 20C0045

Version Date: May 12, 2023 NCT Number: NCT04287868

**RSC Number: 2744** 

Title: Phase I/II Trial of Combination Immunotherapy in Subjects with Advanced HPV

Associated Malignancies

NCI Principal Investigator: Charalampos Floudas, MD, DMSc, MS

Center for Immuno-Oncology (CIO) Center for Cancer Research (CCR) National Cancer Institute (NCI)

10 Center Drive

Building 10, Room 7N240A

Bethesda, MD 20892 Phone: 240-858-3032

Email: <a href="mailto:charalampos.floudas@nih.gov">charalampos.floudas@nih.gov</a>

| Drug Name: | PDS0101 | MSB0011359C<br>(M7824) | NHS-IL12<br>(M9241) |
|---|---|---|---|
| IND Number: | 019267 | 019267 | 019267 |
| Sponsor: | Center for Cancer<br>Research, NCI | Center for Cancer<br>Research, NCI | Center for Cancer<br>Research, NCI |
| Manufacturer: | PDS Biotechnology | EMD Serono, Inc. | EMD Serono, Inc. |
| Supplier: | PDS Biotechnology | EMD Serono, Inc. | EMD Serono, Inc. |

**Commercial Agents:** None


# **PRÉCIS**

## **Background:**

- Metastatic or refractory/recurrent HPV associated malignancies (cervical, anal, oropharyngeal cancers etc.) are poorly palliated by standard therapies. There is an unmet need for active treatments for these tumors.
- In a phase I trial of M7824 (NCT02517398) 15 out of 43 (34.9%) participants with HPV associated malignancies had radiographic tumor responses according to RECIST 1.1 or iRECIST.
- While the response rate observed with M7824 appears to be higher than single agent PD-1 inhibitors alone (15-20%), the majority of patients with these diseases still do not seem to benefit from immunotherapy.
- Preclinical studies suggest that the use of a combination of multiple immunotherapy agents may have improved anti-tumor efficacy.
  - Specifically, preclinical studies have shown that the combination of three immunotherapy agents (1) a therapeutic vaccine against HPV positive cancers (PDS0101), (2) a bifunctional fusion protein targeting PD-L1 and TGF beta (M7824), and (3) a tumor targeted immunocytokine (NHS-IL12) produces greater anti-tumor activity than any single or dual combination of these agents.

## **Objectives:**

• To evaluate the objective response rate (ORR) according to Response Evaluation Criteria (RECIST 1.1) of the combination of (1) a therapeutic vaccine against HPV positive cancers (PDS0101), (2) a tumor targeted immunocytokine (NHS-IL12) and (3) a bifunctional fusion protein targeting PD-L1 and TGF beta (M7824) in subjects with checkpoint naïve advanced HPV associated malignancies.

## **Eligibility:**

- Age  $\geq$  18 years old.
- Subjects with cytologically or histologically confirmed locally advanced or metastatic HPV associated malignancies:
  - o Cervical cancers;
  - o P16+ Oropharyngeal cancers;
  - Anal cancers;
  - o Vulvar, vaginal, penile, and squamous cell rectal cancers;
  - Other locally advanced or metastatic solid tumors (e.g., lung, esophagus) that are known HPV+.
- Prior first line systemic therapy is required unless the participant declines standard treatment after appropriate counseling has been provided.
- Subjects must have measurable disease.


## Design:

- This is a phase I/II trial of combination immunotherapy.
- The trial will be conducted using a Simon optimal two-stage design.
- Participants will receive HPV vaccine + NHS-IL12 + M7824.
- The first six participants will be evaluable for dose limiting toxicities (DLTs) and accrual will only continue to 8 participants who have not been treated with checkpoint inhibitors if less than 2 out of the first 6 participants experience a DLT.
- If three or more out of eight participants who have not been treated with checkpoint inhibitors have objective responses accrual will be expanded to enroll 20 evaluable participants.
- Patients with cervical cancer with prior pelvic radiation and boost brachytherapy will be enrolled in a separate cohort to evaluate safety and preliminary evidence of efficacy.


# **TABLE OF CONTENTS**

| hl | PRÉC | IS | 2 |
|---|---|---|---|
| T. | ABLE | OF CONTENTS | 4 |
| S | ГАТЕ | MENT OF COMPLIANCE | 7 |
| 1. | IN | TRODUCTION | 7 |
| | 1.1 | Study Objectives | 7 |
| | 1.2 | Background and Rationale | 8 |
| 2 | EL | IGIBILITY ASSESSMENT AND ENROLLMENT | . 30 |
| | 2.1 | Eligibility Criteria | . 30 |
| | 2.2 | Screening Evaluation. | . 32 |
| | 2.3 | Participant Registration and Status Update Procedures | . 34 |
| | 2.4 | Baseline Evaluation. | . 35 |
| 3 | ST | UDY IMPLEMENTATION | . 35 |
| | 3.1 | Study Design | . 35 |
| | 3.2 | Drug Administration | . 39 |
| | 3.3 | Study Intervention Compliance | . 40 |
| | 3.4 | Dose Modifications | . 40 |
| | 3.5 | Study Calendar | . 51 |
| | 3.6 | Cost and Compensation. | . 53 |
| | 3.7 | Criteria for Removal from Protocol Therapy and Off Study Criteria | . 53 |
| 4 | CC | DNCOMITANT MEDICATIONS/MEASURES | . 54 |
| | 4.1 | The Following Treatments Should Not Be Administered During the Trial | . 54 |
| 5 | CC | DRRELATIVE STUDIES FOR RESEARCH/PHARMACOKINETIC STUDIES | . 55 |
| | 5.1 | Biospecimen Collection | . 55 |
| | 5.2 | Samples for Genetic/Genomic Analysis | . 57 |
| | 5.3 | Sample Storage, Tracking and Disposition | . 58 |
| 6 | DA | ATA COLLECTION AND EVALUATION | . 60 |
| | 6.1 | Data Collection. | . 60 |
| | 6.2 | Data Sharing Plans | . 61 |
| | 6.3 | Response Criteria | . 61 |
| | 6.4 | Toxicity Criteria | . 68 |
| 7 | NI | H REPORTING REQUIREMENTS / DATA AND SAFETY MONITORING PLAN | . 68 |

| | 7.1 | Definitions | 68 |
|---|---|---|---|
| | 7.2 | OHSRP Office of Compliance and Training / IRB Reporting | 68 |
| | 7.3 | NIH Required Data and Safety Monitoring Plan | 69 |
| 8 | SP | ONSOR PROTOCOL/SAFETY REPORTING | 70 |
| | 8.1 | Definitions | 70 |
| | 8.2 | Assessment of Safety Events. | 71 |
| | 8.3 | Reporting of Serious Adverse Events | 72 |
| | 8.4 | Waiver of expedited reporting to CCR | 72 |
| | 8.5 | Safety Reporting Criteria to the Pharmaceutical Collaborators | 72 |
| | 8.6 | Reporting Pregnancy | 72 |
| | 8.7 | Regulatory Reporting for Studies Conducted Under CCR-Sponsored IND | 73 |
| | 8.8 | Sponsor Protocol Deviation Reporting | 73 |
| 9 | CL | INICAL MONITORING PLAN | 74 |
| 10 | ST | ATISTICAL CONSIDERATIONS | 74 |
| | 10.1 | Statistical Hypothesis | 74 |
| | 10.2 | Sample Size Determination | 75 |
| | 10.3 | Populations for Analyses | 76 |
| | 10.4 | Statistical Analyses | 76 |
| 11 | CC | LLABORATIVE AGREEMENTS | 78 |
| | 11.1 | Cooperative Research and Development Agreement (CRADA) | 78 |
| 12 | Ж | MAN SUBJECTS PROTECTIONS | 78 |
| | 12.1 | Rationale For Subject Selection | 78 |
| | 12.2 | Participation of Children | 78 |
| | 12.3 | Participation of Subjects Unable to Give Consent | 78 |
| | 12.4 | Risks/Benefit Assessment | 79 |
| | 12.5 | Consent Process and Documentation | 80 |
| 13 | RE | GULATORY AND OPERATIONAL CONSIDERATIONS | 82 |
| | 13.1 | Study Discontinuation and Closure | 82 |
| | 13.2 | Quality Assurance and Quality Control | 82 |
| | 13.3 | Conflict of Interest Policy | 82 |
| | 13.4 | Confidentiality and Privacy | |
| 11 | DЦ | ARMACEUTICAL INFORMATION | 83 |


| 14.1 | PDS0101 (IND # 019267) | 83 |
|--------|----------------------------------------|----|
| 14.2 | M7824 (MSB0011359C) (IND # 019267) | 85 |
| 14.3 | NHS-IL12 (IND # 019267) | 89 |
| 15 REF | FERENCES | 91 |
| 16 APP | PENDICIES | 95 |
| 16.1 | Appendix A Performance Status Criteria | 95 |


#### STATEMENT OF COMPLIANCE

The trial will be carried out in accordance with International Conference on Harmonisation Good Clinical Practice (ICH GCP) and the following:

• United States (US) Code of Federal Regulations (CFR) applicable to clinical studies (45 CFR Part 46, 21 CFR Part 50, 21 CFR Part 56, 21 CFR Part 312, and/or 21 CFR Part 812)

National Institutes of Health (NIH)-funded investigators and clinical trial site staff who are responsible for the conduct, management, or oversight of NIH-funded clinical trials have completed Human Subjects Protection and ICH GCP Training.

The protocol, informed consent form(s), recruitment materials, and all participant materials will be submitted to the Institutional Review Board (IRB) for review and approval. Approval of both the protocol and the consent form must be obtained before any participant is enrolled. Any amendment to the protocol will require review and approval by the IRB before the changes are implemented to the study. In addition, all changes to the consent form will be IRB-approved; an IRB determination will be made regarding whether a new consent needs to be obtained from participants who provided consent, using a previously approved consent form.

#### 1. INTRODUCTION

#### 1.1 STUDY OBJECTIVES

## 1.1.1 Primary Objective

• To evaluate the objective response rate (ORR) according to Response Evaluation Criteria (RECIST 1.1) of the combination of (1) a therapeutic vaccine against HPV positive cancers (PDS0101), (2) a tumor targeted immunocytokine NHS-IL12 (M9241) and (3) a bifunctional fusion protein targeting PD-L1 and TGF beta (M7824) in subjects with checkpoint naïve advanced HPV associated malignancies.

## 1.1.2 Secondary Objectives

- To evaluate the safety of the combination of (1) a therapeutic vaccine against HPV positive cancers (PDS0101), (2) a tumor targeted immunocytokine NHS-IL12 (M9241) and (3) a bifunctional fusion protein targeting PD-L1 and TGF beta (M7824) in subjects with advanced HPV associated malignancies.
- To assess progression-free survival time (PFS) according to RECIST 1.1.
- To assess overall survival (OS).
- To assess duration of response and ratio of participants that are hospitalized because of adverse events attributed to disease progression.
- To evaluate the safety of the combination at a reduced dose level in patients with cervical cancer with prior pelvic radiation and boost brachytherapy where a potential higher risk of grade 3 hematuria may exist with the full starting doses of both M7824 and NHS-IL12.

# 1.1.3 Exploratory Objectives

- To conduct exploratory immunologic studies to understand and improve the administered treatment, including:
  - o peripheral immune subset analysis before and on treatment;


o soluble factors circulation (e.g., sCD27 and sCD40 ligand) before and on treatment;

- o tumor tissue immune infiltration before and after treatment.
- To assess responses to therapy using iRECIST.
- To assess responses to therapy by HPV serotype or PD-L1 expression.
- To assess correlation between circulating tumor DNA and response to therapy
- To assess response to therapy in checkpoint refractory disease
- To assess response to therapy by HLA type
- To assess response using reduced doses of NHS-IL12 or M7824

#### 1.2 BACKGROUND AND RATIONALE

## 1.2.1 HPV Associated Malignancies

In the United States, there are more than 30,000 cases of HPV associated cancer annually [1] (Table 1). Metastatic HPV associated malignancies (cervical, anal, oropharyngeal cancers etc.) are often incurable and poorly palliated by standard therapies. Responses to chemotherapy are variable but generally short-lived with median PFS around 3 to 7 months [2-5]. In a Gynecologic Oncology Group randomized trial comparing four cisplatin-based doublets as first line therapy for cervical cancer the response rates were 22-29% and median PFS was 4 to 6 months with median OS 10 to 13 months [6]. The addition of bevacizumab to combination chemotherapy has been reported to increase OS by 3.7 months, but virtually all patients die of their disease within 2 years [7]. Randomized trials of second line therapy are lacking but response rates for single agents are generally reported to be less than 20% [8]. Early evidence suggests that immune checkpoint therapy also has a low response rate in this disease with a phase 1b trial (KEYSTONE 028) showing a 12.5% response rate (3/24 patients) and a phase II study showing a response rate of 13.3% (13/98 patients) to pembrolizumab in patients with recurrent or metastatic cervical cancer [9].

Table 1: Estimated annual incidence of HPV associated cancers in the US

| Site | Incidence of HPV associated cancers | Cases attributed to HPV (%) |
|---|---|---|
| Oropharyngeal | 15,738 | 11,000 (70.1%) |
| Cervix | 11,771 | 10,700 (90.6%) |
| Vulvar | 3554 | 2400 (68.8%) |
| Vaginal | 802 | 600 (75%) |
| Penis | 1168 | 700 (63.3%) |


| Site | Incidence of HPV associated cancers | Cases attributed to HPV (%) |
|---|---|---|
| Rectal (squamous cell) | 750 | 700 (91.1%) |
| Anus | 5,010 | 4,600 (91.1%) |
| Total | 38,793 | 30,700 (79.1%) |

For oropharyngeal cancer, the best estimates of the chemotherapy responsiveness are inferred from looking at the oropharyngeal site in subset analyses from clinical trials for head and neck cancers. In a pivotal clinical trial that established platinum, 5-fluorouracil (5-FU), plus cetuximab as first line therapy in head and neck cancer, patients with oropharyngeal tumors experienced PFS of 4 to 6 months and OS of 8 to 11 months [3]. Immune checkpoint therapy has become the standard second line therapy for metastatic oropharyngeal cancer but response rates are still low with this therapy. As an example, the phase 1b trial (KEYNOTE-012) of pembrolizumab which led to its FDA approval for recurrent or metastatic head and neck squamous cell carcinoma (HNSCC) as second line therapy had a 17.7% response rate (34/192 patients). Response rates were slightly better in HPV positive HNSCC (21.9%) [10], but still occurred in only a minority of the patients.

In regard to metastatic anal cancer, only a handful of randomized trials have been performed in the last 30 years. In the metastatic setting, most of the evidence is limited to small phase II trials, retrospective series, and case reports. A recent retrospective series looking at 77 patients, 44 (55%) of whom received 5-FU in combination with cisplatin, 24 (31%) of whom received carboplatin + paclitaxel, and 11 (14%) of whom received another regimen showed a median PFS of 7 months and median OS of 22 months [5]. As with HNSCC, recent early phase trials evaluating immune checkpoint therapy in this disease have shown that responses here too are limited to around 20% of patients treated. A recent phase II trial of nivolumab for metastatic squamous cell anal cancer showed a 21% response rate (7/33 patients) and a recent phase IB trial (KEYNOTE-028) of pembrolizumab showed a 20% response rate (5/25 patients) [11]. In a recently published phase II trial, Massarelli et al. evaluated the combination of a therapeutic HPV vaccine and Nivolumab [12]. In contrast to previous single therapy immune checkpoint inhibitor trials, they found an overall response rate of 33% showing the potential benefit of Immuno-Oncology (I/O) combination therapy for these diseases.


Table 2 Response in patients treated with ISA101 and Nivolumab (Massarelli JAMA Oncol Sept 27, 2018)

Table 2. Response Overall, in Oropharyngeal Cancer, and by Treatment Historya

| | No. (%) | | | | | |
|---|---|---|---|---|---|---|
| | All Patients<br>(N = 24) | Patients With Oropharyngeal Cancer | | | | |
| Response per RECIST,<br>version 1.1 | | All (n = 22) | Platin-Refractory<br>Disease (n = 17) | Cetuximab-Refractory<br>Disease (n = 8) | Platin- and<br>Cetuximab-Refractory<br>Disease (n = 6) | Received Second-line<br>Treatment (n = 12) |
| Overall response rate | 8 (33) | 8 (36) | 6 (35) | 5 (63) | 3 (50) | 5 (42) |
| Complete response | 2 (8) | 2 (9) | 2 (12) | 1 (13) | 0 | 2 (17) |
| Partial response | 6 (25) | 6 (27) | 4 (24) | 4 (50) | 3 (50) | 3 (25) |
| Stable disease | 3 (13) | 2 (9) | 1 (6) | 0 | 1 (17) | 1 (8) |
| Disease control rateb | 11 (46) | 10 (45) | 7 (41) | 5 (63) | 4 (67) | 6 (50) |
| Progression of disease | 13 (54) | 12 (55) | 10 (59) | 3 (38) | 2 (33) | 6 (50) |

Abbreviation: RECIST, Response Evaluation Criteria in Solid Tumors.

tumors exhibited complete response, partial response, and stable disease and indicates lack of progression per RECIST.

Unfortunately, little data exists evaluating immunotherapy for rarer HPV associated malignancies including metastatic vulvar, vaginal, penile, squamous cell rectal or neuroendocrine cervical cancer.

## 1.2.2 Rationale for Combination of I/O Agents

Preclinical studies are now revealing that an effective immuno-oncology strategy for enhancing anti-tumor responses is the use of multiple immune-mediating agents, each targeting different components of the immune system. These include: (a) induction of an immune response via vaccination directed against tumor-associated antigens, (b) reduction of immunosuppressive entities in the TME by the use of anti-PD1/PDL1 MAb checkpoint inhibitors, and/or reduction of immunosuppressive cytokines such as TGF- $\beta$  with the use of a bifunctional anti-PDL1/TGF- $\beta$ 2 "Trap" designated M7824, and (c) potentiation of the immune response in the TME by the use of the tumor targeting NHS-IL12 immunocytokine.

The LTIB, in collaboration with the GMB, has been able to develop and/or co-develop these agents via a series of CRADAs. Each has been interrogated in a series of preclinical studies and in Phase I/II clinical studies in the CCR as well as by other investigators. Preclinical studies and early clinical studies are demonstrating the relative lack of additional toxicities with enhanced clinical benefit employing combinations of 2 of these agents. Preclinical studies are now demonstrating that the combined use of agents from each of the immune-mediating categories described above elicits the most immune-mediated anti-tumor activities.

#### 1.2.2.1 HPV Vaccine

PDS0101 is a novel nanoparticle-based immunotherapy (therapeutic vaccine) developed to treat genital cancers such as anal, cervical, vulvar cancer etc. and their precancers (late-stage dysplasia/neoplasia), as well as head and neck cancers caused by infection with the human papilloma virus (HPV). PDS0101 is a subcutaneously administered therapy consisting of two vialed components mixed by the investigator at the time of administration. The immunotherapy is composed of liposomal nanoparticles of the pure immunologically active R enantiomer of the

<sup>&</sup>lt;sup>a</sup> Refractory indicates progression of disease within 6 months of treatment.

<sup>&</sup>lt;sup>b</sup> Disease control rate is calculated by adding the percentages of patients whose


cationic (positively charged) lipid DOTAP (dioleoyl-trimethylammonium propane) mixed with 6 lipidated antigenic peptides derived from the HPV-16 E6 and E7 proteins.

In-vivo and in-vitro studies performed in normal and transgenic mouse models as well as in-vitro studies using human lymphocytes in culture demonstrated potent immune modulating effects by R-DOTAP. The pure R stereoisomer of DOTAP acts as a potent activator of the MAP kinase signaling pathway leading to activation and maturation of dendritic cells and subsequent induction of the production and release of cytokines and chemokines critical for promotion of an effective immune response. The positive charge on the surface of R-DOTAP liposomes facilitates their uptake by the dendritic cell. This in turn facilitates uptake of the HPV peptide antigen micelles and the antigenic processing and presentation by dendritic cells to T-cells. The ability of cationic liposomes to destabilize endosomes facilitates antigen delivery into the cytoplasm of the dendritic cells and other antigen presenting cells [13]. Effective induction of cytotoxic T-lymphocyte (CTL) responses and tumor regression has been demonstrated in the pre-clinical studies.



**Figure 1.** Anti-tumor efficacy of DOTAP/E7 vs. CpG-E7 and CFA-E7 in C57BL/6J mice bearing TC-1 HPV+ tumors.

Toxicology studies of R-DOTAP and a prototype R-DOTAP/HPV16-E7 single peptide formulation were evaluated in rats and in non-human primates (monkeys). No deaths or clinical signs related to treatment were observed in any of the studies. No treatment effects on body weight were noted. No treatment-related and/or toxicologically significant effects for any clinical chemistry parameters evaluated were noted during any of the studies. All hematology parameters, red blood cell counts, hemoglobin, mean corpuscular volume, mean corpuscular hemoglobin and mean corpuscular hemoglobin concentration remained normal.

Toxicology of the PDS0101 clinical formulation (6-peptide HPVmix and ImmunoMAPKRDOTAP) was evaluated in humanized transgenic mice. The transgenic mice expressed the human HLA-A2 antigen recognition and presentation molecule, and their antigen presenting cells were therefore capable of recognizing and responding to the HPV A2 epitope human peptide antigens in the drug formulation. Similar to toxicology studies in rats and monkeys


with the prototype drug formulation, few clinically relevant toxicological effects were observed at any dose level in the transgenic humanized mice. However, for the clinical PDS0101 formulation mean hematocrit was decreased in the low R-DOTAP + HPVmix and high R-DOTAP + HPV mix groups by approximately 3% and 5%, respectively; and although minimal, may be related to treatment. No treatment-related toxicological findings were observed during gross necropsy. Microscopic histopathologic findings (minimal fibrosis) considered related to treatment with the test article were limited to the skin at the injection site in 3 out of 8 in the high R-DOTAP + HPV mix group only.

In 2014-2016, a Phase I/IIA human clinical trial was performed at 3 sites in the US in 12 subjects with high-risk HPV infection and biopsy-proven cervical intraepithelial neoplasia (CIN1) to study the safety and immunogenicity of PDS0101. The study initiated with Cohort 1 and progressed through Cohort 3, with each subsequent cohort receiving a higher dose of PDS0101 (i.e., 1.0, 3.0, and 10.0 mg R-DOTAP); 3 in Cohort 1 (1-mg R-DOTAP dose), 3 in Cohort 2 (3 mg R-DOTAP dose), and 6 in Cohort 3 (10-mg RDOTAP dose). Successive cohorts received a constant dose of 2.4 mg HPV-16 E6 and E7 peptides (400 µg/peptide) with 1 of 3 escalating doses of R-DOTAP. All subjects received 3 doses of vaccine given SC, approximately 21 days apart. 10/12 subjects had a positive vaccine-induced response (a  $\geq$ 3-fold increase over baseline at  $\geq$ 1 of the 4 post-vaccination visits by either the IFN- $\gamma$  or granzyme B ELISpot assays, with background counts subtracted). Individual subject results from both the IFN- $\gamma$  and the granzyme B assays showed that all doses of RDOTAP were effective in inducing HPV-specific T-cell responses (Figure 2A). IFN- $\gamma$  (all T-cells) and the granzyme B (CD8+ T-cells) responses were elicited in both HPV-16+ and HPV-16- subjects, and in subjects with various HLA types.

Administration of PDS0101 was also well tolerated. The majority of AEs were due to administration site reactions. Most administration site reactions were mild or moderate in severity. Some more severe administration site reactions including swelling and redness were reported in the 3- and 10-mg R-DOTAP cohorts. Most administration site reactions resolved the same day or within a few days. Per the subject symptoms diary, administration site reactions were more severe and of longer duration in subjects in the 10-mg R-DOTAP cohort. No clinically significant differences in the types and pattern of TEAEs were observed between Vaccinations 1, 2, or 3. No DLTs were observed; thus, the MTD was the 10-mg R-DOTAP dose. No serious adverse events (SAEs), study discontinuations due to adverse events, or deaths occurred. No clinically relevant abnormal hematology, blood chemistry, urinalysis, or physical findings were observed. Regression of CIN was noted in a number of patients (Figure 2B). Regression was seen in CIN related to a variety of HPV types including HPV-16, HPV-18 as well as other high-risk HPV types. The 3-mg R-DOTAP PDS0101 dose (containing 2.7 mg HPV-16 E6 & E7 antigens) has been chosen for further evaluation in larger Phase II trials given it seems to afford the best combination of safety and potency. The original dose of HPV-16 E6 & E7 antigens has been minimally increased from 2.4 mg to 2.7 mg for planned phase II studies. This was done due to some concern with possible oxidation of one of the peptides at the original lower dose. For simplicity the dose of all peptides has been minimally increased.


# Versamune®-HPV (PDS0101) Phase 1 Clinical Trial: Confirmation of unique potential to induce <u>rapid and strong</u> CD4 and CD8 T-cell responses against a viral target (HPV16) <u>14 days post-vaccination</u>



- Strong virus-specific CD8 T-cell responses were also confirmed by Granzyme-b ELISPOT (data not shown)
- · Safe in all subjects: Mild transient vaccine site reactions without systemic toxicity

| | © | , |
|---|---|---|
| Ţ | Versamune®-HPV (PDS0101) Phase 1 Clinical Trial: Regression of CIN Lesions | E |
| <u>_</u> | 0 | -0 |

| Dans Cabart | Evaluable<br>Patients* | Clearance of CIN<br>12 Months Post Treatment** | |
|---|---|---|---|
| Dose Cohort | N = | N = | % of Evaluable |
| 1 mg | 3 of 3 | 2 | 67% |
| 3 mg | 2 of 3 | 1 | 50% |
| 10 mg | 5 of 6 | 3 | 60% |
| Total | 10 | 6 | 60% |

<sup>\*</sup> Two of twelve patients were not evaluable: one patient, who demonstrated a strong immune response (high dose cohort), was lost to follow up and another received standard of care LEEP excision therapy at 4 months (mid dose cohort)

Figure 2 A (top). ELISpot responses in patients treated with PDS0101. B (bottom). CIN Regression in patients treated with PDS0101 [14].

# Avelumab (anti-PD-L1) and M7824 (anti-PD-L1/TGF- βR2)

Studies in the LITB were the first to describe [15, 16] avelumab, a fully human anti-PD-L1 IgG1 MAb, and its ability to mediate ADCC for a range of human carcinoma cells employing NK cells as effectors. Avelumab (Bavencio) has since been approved by the FDA for the therapy of Merkel cell carcinoma (the first drug approved for this indication) and second line urothelial carcinomas. We have also shown that endogenous IL-12 will enhance avelumab-mediated NK lysis, thus

<sup>\*\*</sup> Two of ten evaluable patients who had clearance of CIN by cytology were not considered as clinical responders: one patient regressed from CIN to atypical squamous cells of undetermined significance (ASCUS) with detectable virus, and the other showed consistent disease elimination by cytology, but showed residual disease by colposcopy


forming the basis for the combined use of avelumab or M7824 with NHS-IL12. The first-in-human clinical study of avelumab with over 1,700 patients was led by Gulley with the dose escalation and initial PK and PD done entirely within the CCR [16]. Because of the activity this study was amended to include multiple expansion cohorts internationally. Because PD-L1 is also expressed on some immune cell subsets, our finding [17] that there were no adverse events in the patients treated with avelumab above that seen with other anti-PD-L/PD-L1 MAbs was important for planning further studies with avelumab or M7824.

TGF- $\beta$  is a well-known inhibitor of immune cell function, especially in the TME [18-23]. Prior studies have indicated the advantage in the use of a TGF- $\beta$  inhibitor in combination with checkpoint therapy [24, 25] In collaboration with our CRADA partner EMD Serono, we have supported the development of a bifunctional fusion protein aimed at bringing a TGF- $\beta$  TRAP to tumor cells via binding to PD-L1. M7824 is a novel fusion protein consisting of anti PD-L1 antibody linked to the extracellular domain of two TGF- $\beta$ R2 (serving as a TGF- $\beta$  TRAP) (**Figure 3**).



**Figure 3.** Schematic drawings of Avelumab and M7824.

We were the first to report [26, 27] that M7824 (a) mediates ADCC, (b) increases tumor cell gene expression of molecules involved in T-cell trafficking to the tumor, (c) enhances TRAIL- and antigen-specific CD8+ T-cell lysis of tumor cells, and (d) reduces TGF-β-induced immunosuppressive activity. We have also recently demonstrated [28] in in vivo preclinical murine carcinoma models (Figure 4A and B) that M7824 has the ability to decrease TGF-β-induced signaling in the TME. Specifically, phosphorylation of SMAD2 was significantly decreased in tumors following M7824 treatment, and not with an M7824(mut) molecule, devoid of the PD-L1 binding site (Figure 4C). In both breast and colon carcinoma murine models, M7824 decreased tumor burden and increased survival, which required both CD8+ and NK cell activity (Figure 4D).




**Figure 4 (A)** Comparison of anti-tumor activity of M7824, and M7824(mut) devoid of PD-L1 binding site in the EMT6 breast cancer model. **(B)** Accumulation of M7824 in the TME resulting in reduction of SMAD2 signaling **(C)** and increased T- and NK-cell activation **(D).** Knudson ... Schlom J. OncoImmunology. 2018:e1426519.

Two recent studies [29, 30] demonstrated the advantage in anti-tumor activity in the use of the bifunctional agent vs. the use of a PD- 1/PD-L1 checkpoint in combination with a systemic TGF-β inhibitor. TGF-β is also known to alter human carcinoma cells from a more epithelial to a more mesenchymal phenotype and such tumor cells are more resistant to a range of therapies (**Figure 5**). In LTIB studies, TGF-β-induced mesenchymalization of carcinoma cells was shown [31] to be reversed by M7824, rendering tumor cells more susceptible to chemotherapy and immune-mediated killing [26, 28, 31]

The first-in-human trial of M7824 (anti-PD-L1/TGF- $\beta$ R2) was conducted at the CCR [32]. Nineteen heavily pretreated patients with solid tumors (non-melanoma) were treated; the MTD was not reached. M7824 was shown to saturate peripheral PD-L1 and sequester all released (acid released) plasma TGF $\beta$ 1, - $\beta$ 2, and - $\beta$ 3 throughout the dosing period at >1 mg/kg (recommended phase 2 dose is 1200 mg or about 10 mg/kg). There were signs of clinical efficacy across all dose levels (Figure 6 and Figure 7), including one ongoing CR (cervical cancer), two durable PRs (pancreatic and anal cancers), one near PR (cervical) and two cases of prolonged stable disease.




**Figure 5.** Functions of M7824.




**Figure 6.** Phase I trial of M7824, spider plot of tumor responses and reduction of serum levels of TGFβ1.




Figure 7. M7824 Phase I, responses in two patients.

In the Phase I study [32] 15/43 (34.9%) of patients with checkpoint naïve HPV associated malignancies had radiographic tumor responses according to RECIST 1.1 or iRECIST with M7824 (anti-PD-L1/TGF- $\beta$ R2) therapy. Prior studies by others have shown approximately a 15% objective response in this population employing checkpoint inhibition therapy. In an ongoing phase II study (NCT03427411) 3/22 (13.6%) patients with checkpoint refractory advanced HPV associated malignancies have had responses to M7824 which compares well to the less than 5% response rate seen in the literature with further checkpoint therapy.

Sufficient peripheral blood mononuclear cells were available from 12 patients on the phase I trial to test for HPV-specific T-cell responses before and after M7824 treatment. Considering all post-therapy timepoints examined, 7 of 12 patients (58%) had an increase in HPV-specific T cells post-vs pre-M7824 therapy. Immune responses after 1 and 3 cycles of M7824 were compared between patients who developed a clinical response of stable disease or better vs those with progressive disease (Figure 8). In clinical responders, HPV-specific T cells developed in 3 of 4 patients (75%) after 1 cycle of M7824 and in 4 of 4 patients (100%) after 3 cycles. On the other hand, in patients with progressive disease, HPV-specific T cells developed in only 1 of 5 patients (20%) after 1 cycle of M7824 and in 1 of 4 patients (25%) after 3 cycles (Supplementary Table 3). There was also an increased magnitude of HPV-specific T cells generated in clinical responders vs


nonresponders: clinical responders had on average 12- to 27-fold more HPV-specific T cells producing cytokines or positive for CD107a (LAMP1, a functional marker of T and NK cell activity) after 1 and 3 cycles of M7824 compared with nonresponders (Figure 3A).

Another observation worth noting is that 2 of the 3 patients with HPV+ cancer who received prior lymphodepleting chemotherapy (e.g., cyclophosphamide, fludarabine) were assessed for immune responses post- vs pre-M7824 therapy, and neither had evidence of an HPV T-cell–specific immune response. In contrast, in patients with HPV+ cancer who did not receive prior lymphodepleting chemotherapy, 6 of 9 (67%) had a positive T-cell–specific immune response.



**Figure 8.** Immune responses in HPV+ patients with disease control (BOR of SD, PR, or CR) vs nonresponders (BOR of PD) to M7824 therapy by intracellular cytokine staining following in vitro stimulation with a mixture of overlapping 15-mer peptide pools encoding HPV-16 E6 and E7, as previously described.<sup>21</sup>


## NHS-IL12 Immunocytokine (M9241)

NHS-IL12 is a tumor targeting immunocytokine that binds to DNA-histone in necrotic areas of tumor. Studies by others have shown the ability of radiolabeled NHS-IL12 to target murine and human tumors (**Figure 9**). Prior studies in the LTIB have shown the ability of this agent to elicit anti-tumor activity in multiple murine models, and in combination with anti-PD-L1 and with radiation and chemotherapy [33]. Gulley (GMB, CCR) and the LTIB conducted the Phase I dose escalation trial of the NHS-IL12 immunocytokine [34]. Due to known prior toxicities using a rec.



**Figure 9.** NHS-IL12 Immunocytokine. **(A)** NHS76 is a fully human 2<sup>nd</sup> generation TNT antibody bound to 2 murine IL-12 (p70) molecules. **(B) a:** Specific tumor targeting of transplanted lung carcinoma by the MAb NHS-IL12(mu). Control MAb BC1-IL12(mu). **b:** NHS-IL12 tumor targeting of nuclear DNA histones.

IL-12 protein, multiple ascending dose levels were employed and the agent was administered every 4 weeks. Time-dependent increase in serum IFN-γ and subsequent rise in IL-10 increased with dose and varied greatly among patients (**Figure 10A**). Increases in TCR diversity and TIL density in the TME following NHS-IL12 dosing were observed in those patients with elevation IFN-γ serum levels (**Figure 10B**). Toxicity was acceptable with an MTD of 16.8 mcg/kg and this total dose was also found to be safe when given split in half on an every 2 week schedule. Although no objective tumor responses were seen, of 30 patients with measurable disease, 15 had stable disease, with some durable (from 6–30+ months).




**Figure 10. (A)** Diversity of IFN-γ spikes in sera among patients 3 days post-NHS-IL12 treatment for cycles 1 (C1) and 2 (C2): as examples, 2 patients with high (pts 1 and 2, red and blue) and low (pts 3 and 4, green and orange) levels are shown. **(B)** Changes in TCR clonal diversity in the tumor biopsy correlate with serum IFN-g responses post-NHS-IL12 treatment. **(C)** # of clones in tumor comprising the top 25% of the repertoire of patient 1 pre- and post-NHS-IL12, demonstrating an increase in TCR diversity in a high IFN-g responder after therapy.


Our recent preclinical studies have also shown the enhanced anti-tumor effect of avelumab when used in combination with NHS-IL12 in syngeneic mice bearing an intravesical bladder tumor (Figure 11, left panel) and that this effect is mediated via an IFN- $\gamma$ -dependent mechanism. Studies in NSG- $\beta$ 2m<sup>-/-</sup> mice bearing HTB1, a human bladder carcinoma, and reconstituted with human PBMC, also showed the enhanced anti-tumor effect of the combination that coincided with increased NK and CD8<sup>+</sup> in the TME (Figure 11, right panel).



**Figure 11.** Anti-tumor activity of NHS-IL12 + anti-PD-L1 in NSG-β2m<sup>-/-</sup> mice bearing human bladder cancer (HTB1).

This further provided the rationale for an ongoing CCR led clinical study of avelumab in combination with NHS-IL12 (NCT02994953), currently evaluating safety of the combination. In addition, to the combination being found to be safe and well-tolerated, evidence of radiographic tumor responses has been observed. As an example, a patient with checkpoint refractory metastatic urothelial cancer with a large sacral mass and retroperitoneal adenopathy at enrollment has had an ongoing complete response for 18+ months.

#### **Combination Immunotherapies**

In addition to harnessing the potential multi-functionality of M7824, we have conducted several combination studies employing this agent with other immune modulating agents. We have previously shown [27] enhanced anti-tumor activity when M7824 was combined with vaccine in EMT6, a metastatic breast carcinoma murine model (Figure 12).




**Figure 12.** Combined effect of Ad-Twist vaccine and M7824 in EMT6 breast carcinoma model (Knudson, 2018)

Furthermore, combining M7824 with NHS-IL12 also greatly enhanced anti-tumor activity in the EMT6 breast carcinoma model (Figure 13). Tumor challenge studies showed the presence of immune memory in mice that received the combination of M7824 and NHS-IL12, which conferred protection against re-challenge with tumor. Similar results were also seen in the MB38-CEA murine colorectal carcinoma model.



Figure 13. Anti-tumor effect of M7824 + NHS-IL12 combination treatment in EMT6.

Multimodal therapies were also carried out in mice bearing HPV<sup>+</sup> tumors. The combination of PDS0101 vaccine and M7824 showed significant anti-tumor efficacy in the NSG  $\beta$ 2m<sup>-/-</sup>humanized mouse model reconstituted with human PBMC and bearing human cervical HPV<sup>+</sup> cancer (SiHa) subcutaneously (**Figure 14**).




| Treatment | Tumor volume<br>>200 mm <sup>3</sup> |
|---------------|--------------------------------------|
| PBS Control | 6/12 |
| M7824 | 4/12 |
| PDS0101 | 5/12 |
| PDS0101+M7824 | 1/12 |

**Figure 14.** Tumor growth in humanized mice bearing SiHa (human HPV<sup>+</sup> cervical cancer) and treated with PBS control, PDS0101 vaccine, M7824, or PDS0101+M7824.

In contrast to the previous clinical trials, where we saw anti-tumor efficacy of M7824 or PDS0101 alone in HPV-associated tumors, in this model there was no single therapy effect of M7824 or PDS0101, but the combination significantly decreased tumor burden. Furthermore, in C57BL/6J mice bearing TC-1 (a murine lung carcinoma line transfected with HPV16 E6 and E7 oncoproteins), which is a very aggressive model of HPV<sup>+</sup> carcinoma, the combination of PDS0101 vaccine, M7824 and NHS-IL12 resulted in the greatest level of anti-tumor activity compared to the use of individual agents or dual combinations (Figure 15). The use of the combination of PDS0101 vaccine, M7824 and NHS-IL12 also resulted in an intense influx of CD4<sup>+</sup> and CD8<sup>+</sup> T cells in tumors (Figure 16, upper panels and Figure 17), increased activation and proliferation of T-cells (Figure 16, lower panels), as well as an enhanced HPV specific T cell response measured by ELISpot not seen with lesser combinations (Figure 18).




**Figure 15 A.** Tumor growth in C57BL/6J mice bearing TC-1 HPV+ tumors, and treated with combinations of PDS0101, M7824, and NHS-IL12.

| Treatment | Tumor Volume<br><300mm <sup>3</sup> |
|-------------------|-------------------------------------|
| PBS Control | 0/16 |
| DOTAP | 0/8 |
| M7824 | 0/16 |
| PDS0101 | 3/16 |
| NHS | 6/16 |
| M7824+NHS | 8/16 |
| PDS0101+NHS | 10/16 |
| PDS0101+M7824 | 5/16 |
| PDS0101+M7824+NHS | 13/17 |

**Figure 15 B.** Tumor control (low volume) in C57BL/6J mice bearing TC-1 HPV+ tumors, and treated with combinations of PDS0101, M7824, and NHS-IL12.



**Figure 16.** Increased T-cell infiltration by tumor weight, and increased T-cell activation and proliferation in combination treated mice. (Rumfield et al; unpublished)


# Immunohistochemistry for CD4+ and CD8+



**Figure 17.** Immunohistochemistry shows increased T-cell infiltration in C57BL/6J mice bearing TC-1 HPV+ tumors, and treated with the combination of PDS0101, M7824, and NHS-IL12.


## **HPV 16 E7 15-mer**



| Treatment | Tumor Volume<br><300mm <sup>3</sup> | E7 ELISpot |
|-------------------|-------------------------------------|------------|
| PBS Control | 0/16 | - |
| DOTAP | 0/8 | - |
| M7824 | 0/16 | - |
| PDS0101 | 3/16 | + |
| NHS | 6/16 | - |
| M7824+NHS | 8/16 | - |
| PDS0101+NHS | 10/16 | + |
| PDS0101+M7824 | 5/16 | + |
| PDS0101+M7824+NHS | 13/17 | - |

**Figure 18.** PDS0101 generated HPV-specific T-cells, as measured by ELISpot. Table shows a summary of tumor volume and E7-specific IFNγ ELISpot for C57BL/6J mice bearing TC-1 HPV+ tumors, and treated with combinations of PDS0101, M7824, and NHS-IL12

## 1.2.3 Safety and Efficacy of I/O Combinations in Humans

**Table 3:** Previously evaluated combinations of I/O agents demonstrating an acceptable safety profile.

| Avelumab (anti-PD-L1) + NHS-IL12 | NCT02994953 |
|----------------------------------|-------------|
| CEA/ MUC1 vaccine + M7824 | NCT03315871 |

Dose Rationale: In the phase I dose escalation trial of combination Avelumab (anti-PD-L1) + NHS-IL12, escalating doses of NHS-IL12 were evaluated at 8,12, and 16.8 mcg/kg given every 4 weeks in combination with standard dosing of Avelumab. The combination including NHS-IL12 at the highest dose evaluated (16.8 mcg/kg given every 4 weeks) was found to be well tolerated. The only DLT observed on the trial was a transient grade 3 AST/ALT elevation at NHS-IL12 at 12 mcg/kg but otherwise no other DLT was observed and the MTD was not reached. Therefore,


for this protocol, NHS-IL12 was originally used at a dose of 16.8 mcg/kg every 4 weeks in combination with the standard phase II dose of M7824 of 1200 mg given every two weeks. While we observed no DLTs with the combination of NHSIL12 at 16.8 mcg/kg along with M7824 and PDS0101 in the six participant lead in safety cohort, after treating 19 participants on protocol we observed that the majority of participants (11/19; 57.9%) needed dose reductions of NHSIL12 when given in combination with PDS0101 and M7824 due mostly to grade 2 fever and flu like symptoms.

At this point (with Protocol Amendment Version 12.11.2020) we lowered the starting dose of NHS-IL12 in this protocol from 16.8 mcg/kg to 8 mcg/kg to try and minimize toxicity. After evaluating a total of 39 patients on this protocol including 21 with starting dose of 16.8 mcg/kg and 18 patients with starting dose of 8 mcg/kg we observed what looks to be reduced efficacy in patients receiving 8 mcg/kg as a starting dose with only 3/18 patients responding with the 8 mcg/kg starting dose as compared to 11/21 with the 16.8 mcg/kg starting dose. Therefore, based on this observation that the possibility that a lowering starting dose of NHS-IL12 may reduce efficacy we are amending to allow treatment (effective with Protocol Amendment Version 09.20.2021) with a limited number of doses of NHS-IL12 at 16.8 mcg/kg (four doses total), followed by dosing at 8 mcg/kg every 4 weeks thereafter. This is based upon responding patients in the first 21 patients which received anywhere between 1-4 doses of NHS-IL12 at 16.8 mcg/kg before dose reductions.

## 1.2.4 Immune Assays

Multiple immune assays have been developed in the LTIB to better define the mechanism(s) involved in the use of specific novel agents, as monotherapy or in combination therapies, both for preclinical and clinical studies. In addition to analyses of biopsies, analyses of the peripheral immunome can provide valuable information in that multiple samples can be analyzed over the course of a given therapy vs. pre-therapy. The LTIB has now developed and employed [15, 16, 31, 35] a flow cytometry–based assay that can analyze 123 immune cell subsets in human PBMC from one vial of processed PBMC (approximately 107 cells). This assay will be used in this clinical trial to detect multiple (n=32) subsets of CD4+ T cells, CD8+ T cells (n=29), Tregs (n=7), B cells (n=5), NK (n=20), NKT (n=4), DC (n=10), and MDSC (n=16) to better understand the role of each agent. We also plan to evaluate changes in TCR clonal diversity both in biopsies and the periphery. One example involves an ongoing first-in-human trial of the NHS-IL12 tumor-targeting immunocytokine. TCR diversity increased 6-14-fold in biopsies of patients with a high or intermediate IFN-y response but were unchanged or decreased with a low IFN-y response. These findings also correlated with TIL in biopsies. We are also currently employing NanoString analyses to identify a gene signature in biopsies and PBMC, pre- and post-treatment. The GMB will conduct multiplexed, multispectral imaging of FFPE tissue to evaluate multiple immune parameters within the TME before and after treatment in patients with available tissue.

#### 1.2.5 Summary

- We are proposing a novel I/O combination to help overcome multiple barriers in an effective anti-tumor immune response.
  - o (1) HPV therapeutic vaccine targeting tumor associated antigens to prime an antitumor immune response
  - o (2) NHS-IL12 and M7824 to enable activated immune cells to work better in the TME


 Preclinical studies have shown that treatment with the combination of an HPV therapeutic vaccine, M7824 and NHS-IL12 leads to greater anti-tumor activity than any single or double combination of these agents

#### 2 ELIGIBILITY ASSESSMENT AND ENROLLMENT

#### 2.1 ELIGIBILITY CRITERIA

- 2.1.1 Inclusion Criteria
- 2.1.1.1 Subjects with cytologically or histologically confirmed locally advanced or metastatic HPV associated malignancies:
  - Cervical cancers;
  - P16+ Oropharyngeal cancers;
  - Anal cancers;
  - Vulvar, vaginal, penile, and squamous cell rectal cancers;
  - Other locally advanced or metastatic solid tumors (e.g., lung, esophagus) that are known HPV+.
- 2.1.1.2 Subjects must have measurable disease, per RECIST 1.1. See Section 6.3 for the evaluation of measurable disease.
- 2.1.1.3 Subjects must have received one prior line of systemic chemotherapy as well as checkpoint therapy if checkpoint therapy is FDA approved for that specific tumor type (e.g., HNSCC and PDL1+ cervical cancer). Prior checkpoint therapy is not needed where checkpoint therapy has not been FDA approved for that specific tumor type (e.g. anal, vaginal, vulvar, penile, PDL1 negative cervical). Exceptions to the above include participant who are not eligible to receive the above therapies or who decline these standard treatment options after appropriate counseling has been provided.
- 2.1.1.4 Age >18 years.
- 2.1.1.5 ECOG performance status < 2.
- 2.1.1.6 Adequate hematologic function at screening, as follows:
  - Absolute neutrophil count (ANC)  $\geq 1 \times 10^9/L$ ;
  - Hemoglobin  $\geq 9 \text{ g/dL}$ ;
  - Platelets  $\geq 75,000/\text{microliter}$ .
- 2.1.1.7 Adequate renal and hepatic function at screening, as follows:
  - Serum creatinine ≤ 1.5 x upper limit of normal (ULN) OR
     Measured or calculated creatinine clearance ≥ 40 mL/min for participant with
     creatinine levels > 1.5 X institutional ULN (GFR can also be used in place of
     creatinine or CrCl);
  - Bilirubin  $\leq 1.5$  x ULN OR in subjects with Gilbert's syndrome, a total bilirubin  $\leq 3.0$  x ULN:
  - Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)  $\leq$  2.5 x ULN, unless liver metastases are present, then values must be  $\leq$  3 x ULN).
- 2.1.1.8 The effects of the immunotherapies on the developing human fetus are unknown. For this reason and because immunotherapeutic agents as well as other therapeutic agents used in


this trial are known to be teratogenic, women of child-bearing potential and men must agree to use highly effective contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for two months after study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

- 2.1.1.9 Participants serologically positive for HIV, Hep B, Hep C are eligible as long as the viral loads are undetectable by quantitative PCR. HIV positive participants must have CD4 count ≥ 200 cells per cubic millimeter at enrollment, be on stable antiretroviral therapy for at least 4 weeks and have no reported opportunistic infections or Castleman's disease within 12 months prior to enrollment.
- 2.1.1.10 Ability of subject to understand and the willingness to sign a written informed consent document.

#### 2.1.2 Exclusion Criteria

- 2.1.2.1 Participants with prior investigational drug, chemotherapy, immunotherapy or any prior radiotherapy (except for palliative bone directed therapy) within the past 28 days prior to the first drug administration except if the investigator has assessed that all residual treatment-related toxicities have resolved or are minimal and feel the participant is otherwise suitable for enrollment. Participants may continue adjuvant hormonal therapy in the setting of a definitively treated cancer (e.g., breast cancer).
- 2.1.2.2 Known intolerance to or life threatening side effects resulting from prior checkpoint inhibitor therapy.
- 2.1.2.3 Major surgery within 28 days prior to the first drug administration (minimally invasive procedures such as diagnostic biopsies are permitted).
- 2.1.2.4 Known active brain or central nervous system metastasis (less than a month out from definitive radiotherapy or surgery), seizures requiring anticonvulsant treatment (<3 months) or clinically significant cerebrovascular accident (<3 months). In order to be eligible participants must have repeat CNS imaging at least a month after definitive treatment showing stable CNS disease. Participants with evidence of intratumoral or peritumoral hemorrhage on baseline imaging are also excluded unless the hemorrhage is grade ≤ 1 and has been shown to be stable on two consecutive imaging scans.
- 2.1.2.5 Pregnant women are excluded from this study because these drugs have not been tested in pregnant women and there is potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these immunotherapies, breastfeeding should be discontinued if the mother is treated on this protocol.
- 2.1.2.6 Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent with exception of:
  - Diabetes type I, eczema, vitiligo, alopecia, psoriasis, hypo- or hyperthyroid disease or other mild autoimmune disorders not requiring immunosuppressive treatment;
  - Subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses ≤ 10 mg of prednisone or equivalent per day;


• Administration of steroids for other conditions through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) is acceptable;

- Subjects on systemic intravenous or oral corticosteroid therapy with the exception of physiologic doses of corticosteroids (≤ the equivalent of prednisone 10 mg/day) or other immunosuppressives such as azathioprine or cyclosporin A are excluded on the basis of potential immune suppression. For these subjects these excluded treatments must be discontinued at least 1 weeks prior to enrollment for recent short course use (≤ 14 days) or discontinued at least 4 weeks prior to enrollment for long term use (> 14 days). In addition, the use of corticosteroids as premedication for contrast-enhanced studies is allowed prior to enrollment and on study.
- 2.1.2.7 Subjects with a history of serious intercurrent chronic or acute illness, such as cardiac or pulmonary disease, hepatic disease, bleeding diathesis or recent (within 3 months) clinically significant bleeding events, or other illness considered by the Investigator as high risk for investigational drug treatment.
- 2.1.2.8 Subjects unwilling to accept blood products as medically indicated.
- 2.1.2.9 History of non-HPV associated second malignancy within 3 years of enrollment except localized malignancy which has been adequately treated or malignancy which does not require active systemic treatment (e.g., low risk CCL). Patients taking adjuvant hormonal therapy for definitively treated cancers (e.g. breast cancer) are eligible.
- 2.1.2.10 Subjects with a known severe hypersensitivity reaction to a monoclonal antibodies (grade >/= 3 NCI-CTCAE v5) will be evaluated by the allergy/immunology team prior to enrollment.
- 2.1.2.11 Receipt of prior lymphodepleting chemotherapy (e.g. cyclophosphamide, fludarabine) or any organ transplantation requiring ongoing immunosuppression.

## 2.1.3 Recruitment Strategies

This study will be posted on <a href="www.clinicaltrials.gov">www.clinicaltrials.gov</a>, NIH websites and on NIH social media forums. After IRB approval of the recruitment material, this study may be advertised at national conferences including AACR and ASCO and may also be shared with the HPV and Anal Cancer Foundation who may advertise it further.

Participants will be recruited from the current participant population at NIH. Participants with HPV related cancers are currently being treated on another trial through LTIB, CCR, NIH, where 2-3 participants per month are being screening and enrolled. Some of these participants come from established community networks, some of these participants are self-referrals, and some of these participants are referred by another group (Dr. Hinrichs's group, ETIB, CCR, NIH) who also have a large referral base for HPV related cancers.

#### 2.2 SCREENING EVALUATION

2.2.1 Screening activities prior to the obtaining informed consent

Minimal risk activities that may be performed before the subject has signed a consent include the following:

• Email, written, in person or telephone communications with prospective subjects


- Review of existing medical records to include H&P, laboratory studies, etc.
- Review of existing MRI, x-ray, or CT images
- Review of existing photographs or videos
- Review of existing pathology specimens/reports from a specimen obtained for diagnostic purposes

## 2.2.2 Screening activities performed after a consent for screening has been signed

The following activities will be performed only after the subject has signed the study consent or the consent for study # 01C0129 (provided the procedure(s) are permitted on that study) on which screening activities will be performed. Assessments performed at outside facilities or on another NIH protocol within these timeframes below may also be used to determine eligibility once a participant has signed the consent.

Within 28 days prior to enrollment, unless otherwise specified:

- Complete medical history and physical examination (including height, weight, vital signs, and ECOG performance status).
- CT of chest, abdomen and pelvis.
- A brain CT scan in participants with known CNS disease as described in Section 2.1.2.4.
- For skin lesions, documentation by color photography, including a ruler to estimate the size of the lesion.
- EKG
- Clinical laboratory tests (within 16 days prior to enrollment).
  - Chemistry: sodium, potassium, chloride, bicarbonate, calcium, glucose, BUN, creatinine, ALT, AST, alkaline phosphatase, total protein, albumin, and total and direct bilirubin.
  - Hematology: complete blood count (CBC) with differential.
  - CD4 (if clinically indicated).
  - HLA typing (where feasible)
- Urine or serum pregnancy test ( $\beta$ -HCG) for females of childbearing-potential and women < 12 months since the onset of menopause (within 16 days prior to enrollment).
- Urinalysis.
- HBV, HCV, HIV testing including viral load if clinically indicated (within 3 months prior to enrollment).
- Histologic confirmation (at any time point prior to enrollment). If there is no available tumor sample or pathology report, a biopsy will be performed to confirm the diagnosis.


## 2.3 PARTICIPANT REGISTRATION AND STATUS UPDATE PROCEDURES

Registration and status updates (e.g., when a participant is taken off protocol therapy and when a participant is taken off-study) will take place per CCR SOP ADCR-2, CCR Participant Registration & Status Updates found at: <a href="https://ccrod.cancer.gov/confluence/pages/viewpage.action?pageId=73203825">https://ccrod.cancer.gov/confluence/pages/viewpage.action?pageId=73203825</a>.

#### 2.3.1 Screen Failure

Screen failures are defined as participants who consent to participate in the clinical trial but are not subsequently assigned to the study intervention or entered in the study. A minimal set of screen failure information is required to ensure transparent reporting of screen failure participants, to meet the Consolidated Standards of Reporting Trials (CONSORT) publishing requirements and to respond to queries from regulatory authorities. Minimal information includes demography, screen failure details, eligibility criteria, and any serious adverse event (SAE).

Individuals who do not meet the criteria for participation in this trial (screen failure) because of a transient lab abnormality may be rescreened.

## 2.3.2 Treatment Assignment Procedures

#### Cohorts

| Number | Name | Description |
|---|---|---|
| 1 | Cohort 1 | Subjects with HPV associated malignancies |
| 2 | Cohort 2 | Subjects with cervical cancer with prior pelvic radiation and boost brachytherapy |

2

#### Arms

| Number | Name | Description |
|--------|-------|-------------------------------------------------|
| 1 | Arm 1 | HPV vaccine + NHS-IL12 + M7824 |
| 2 | Arm 2 | HPV vaccine + NHS-IL12 + M7824 at reduced doses |

## **Arm Assignment**

Participants in Cohort 1 will be assigned to Arm 1, and patients in Cohort 2 will be assigned to Arm 2. If more than three of eight patients have an objective response then accrual will be expanded to enroll 20 evaluable participants for cohort 1, while cohort 2 may enroll up to 12 patients for a safety evaluation and up to 12 additional patients for preliminary evaluation of efficacy as well as further evaluation of safety


#### 2.4 BASELINE EVALUATION

All subjects are required to complete baseline evaluations within one week prior to the first planned dosing of the study drug (any screening evaluation done within this time period can also serve for the baseline evaluation):

- Physical exam including weight, ECOG performance status and vital signs.
- Concomitant Medications and Baseline Signs and Symptoms evaluation.
- Urine or serum pregnancy test ( $\beta$ -HCG) for females of childbearing-potential and women < 12 months since the onset of menopause.
- Chemistry: sodium, potassium, chloride, bicarbonate, calcium, glucose, BUN, creatinine, ALT, AST, alkaline phosphatase, total protein, albumin, and total and direct bilirubin.
- ACTH, TSH, reflex free T4, lipase, amylase, CRP
- Hematology: CBC with differential
- Coagulation panel: PT, INR, and PTT

#### 3 STUDY IMPLEMENTATION

## 3.1 STUDY DESIGN

- This is a phase I/II trial of combination immunotherapy.
- The trial will be conducted using a Simon optimal two-stage design.
- Participants will receive HPV vaccine + NHS-IL12 + M7824 (Figure 19).
  - The first six participants will be evaluable for dose limiting toxicities (DLTs) and accrual will continue to 8 participants if less than 2 out of the first 6 participants experience a DLT.

If three or more out of eight patients have objective responses then accrual will be expanded to enroll 20 evaluable participants (Figure 20). Additional patients will be enrolled in the cohort with prior pelvic radiation and boost brachytherapy: up to 12 for safety and dose finding and up to 12 for an exploratory evaluation of efficacy.

- There will be a minimum of six days between the first and second participant. The third through sixth participant may enroll no sooner than 48 hours after the most recent enrollee. Once six participants have enrolled and been found to be safe further participants may enroll at any time.
- Although positive HPV testing will not be required prior to enrolling, HPV testing will be
  offered as an exploratory endpoint and participants testing negative for HPV after enrolling
  or whose HPV status cannot be confirmed may be replaced with other participants for the
  primary efficacy analysis. Participants testing negative for HPV after enrolling or whose
  HPV status cannot be confirmed may continue to receive treatment on study.
- The combination of PDS0101+ NHS-IL12+ M7824 will be evaluated in all HPV serotypes given the clinical remissions PDS Biotechnology has observed in CIN studies with PDS0101 in non-HPV 16 serotypes. However, if it is found that the ORR with non-HPV-


16 serotypes is noticeably less than the ORR observed with HPV 16 serotypes than participants having disease related to non-HPV-16 serotypes may be replaced with participants having disease related to the HPV-16 serotype for the first and second stage of the primary efficacy analyses.

- In addition, while the primary focus of this protocol is to evaluate the response rate of this I/O combination in participants with a wide array of HPV associated malignancies, if the I/O combination in not deemed to be promising in this larger population (less than three out of eight evaluable participants have a response) than the study will be amended to evaluate this I/O combination specifically in participants with cervical cancer (and participants who have already been enrolled with non-cervical cancers may be replaced with cervical cancer participants for the first stage of the primary efficacy analyses).
- While checkpoint refractory participants will be eligible to enroll, the primary objective of response rate will be determined among the checkpoint naïve participants and the response rate among checkpoint refractory participants will be an exploratory objective.


Figure 19.



Figure 20.


# 3.1.1 Dose Limiting Toxicity

## **DLT** for first 6 participants:

Dose-limiting toxicity (DLT) will be defined as any one of the following adverse events, possibly attributable to study drugs, that occur within 28 days of the start of therapy:

- Any Grade 4 or higher adverse drug reactions (ADRs) as defined by CTCAE v5.0 and assessed as possibly related to that agent by the Investigator, except for laboratory values that are asymptomatic or resolve to Grade ≤ 1 or baseline grade within 7 days without medical intervention.
- Any Grade 3 ADRs possibly attributed to an agent except for any of the following:
  - Grade 3 flu-like symptoms or fever, as well as associated symptoms of fatigue, headaches, nausea, emesis which can be controlled with conservative medical management.
  - O Tumor flare phenomenon defined as local pain, irritation, or rash localized at sites of known or suspected tumor.
  - Grade 3 Hgb decrease (< 8.0 g/dL) that is clinically manageable with blood transfusions or erythroid growth factor use does not require treatment discontinuation.
  - o Grade 3 laboratory values that are asymptomatic or resolve to Grade  $\leq 1$  or baseline grade within 14 days.
  - o Keratoacanthoma and squamous cell carcinoma of the skin.
  - o Any endocrinopathy that can be medically managed with hormone replacement
  - O Any grade 3 adverse drug reaction which can be medically managed with minimal risk to the participant (e.g., placement of a pleural catheter for recurrent inflammatory pleural effusions) and resolves to at least grade one or baseline grade within 14 days.

Criteria are based on the NCI Common Terminology Criteria for Adverse Events, Version 5.

Where clinically appropriate subjects will receive one year of treatment during which subjects will be followed with surveillance scans every 6-12 weeks. On a case by case basis treatment beyond a year is allowed per investigator discretion. Subjects with evidence of disease progression after completing a year of treatment will be allowed retreatment.

Patents might be taken off treatment for disease progression prior to completing one year of treatment, but where clinically appropriate, treatment beyond radiographic progression is allowed if in the opinion of the investigator the subject is benefiting from treatment.

Subjects will be taken off treatment if unacceptable toxicity occurs and is attributed to all therapeutic agents. If a single agent is tolerated that agent may be continued.

This trial will be conducted using a Simon two-stage phase II trial design in which 8 evaluable participants will enroll and if 3 or more of the 8 have an objective response, then accrual would continue until a total of 20 evaluable participants have been treated. If there are 9 or more of 20 (45.0%) who experience a response, this would be sufficiently interesting to warrant further study.

In the event that a participant develops a response (>30% decrease in target lesions as compared with baseline scan) following initial progression or "pseudo-progression", this response will be considered as an objective response in the determination to expand accrual.


#### 3.2 DRUG ADMINISTRATION

#### **General Rule:**

A window of +/- 14 days for a scheduled treatment is allowed in the event of scheduling issues (i.e., holiday, bad weather or other scheduling issues). The minimum time between administrations of a similar agent is 11 days. Where feasible PDS0101 should be administered first, followed by NHS-IL12 (when given), followed by M7824.

#### 3.2.1 PDS0101

PDS0101 will be administered every 4 weeks for 6 doses followed by every three months (i.e. every 12 weeks) for an additional two doses.

Dosage Form: Sterile injectable liquid

Number of vials: 2-vial formulation

Preparation: 1:1 v/v mixture of the 2 vial formulation. 0.6mL of vial #1,

ImmunoMAPK-RDOTAP added to vial# 2, HPVmix (0.6

mL)

Total Administered

dose:

2.7 mg of total peptide and 3 mg of R-DOTAP

Total Injection Volume: 1.0mL (administered as two individual 0.5mL injections)

Injection route: Subcutaneous

• 0.6 ml will be drawn up from each vial (Vial #1 Immuno MAPK-RDOTAP, Vial #2 HPV mix) and mixed (total = 1.2ml for the PDS0101 admixture). Two separate 0.5 ml doses will be injected into the participant. These should preferably be given ~6cm apart in the same limb. Each subsequent vaccination should preferably be administered alternating between limbs (e.g., L arm → R thigh).

#### 3.2.2 M7824

Subjects will receive M7824 via IV infusion over 1 hour (-10 minutes / +20 minutes, that is, over 50 to 80 minutes) once every 2 weeks. M7824 will be administered as a "flat" dose of 1,200 mg independent of body weight. However lower doses may also be used as per Section 3.4.3. M7824 is administered as an intravenous infusion with a mandatory 0.2 micron in-line filter.

In order to mitigate potential infusion-related reactions, premedication with an antihistamine and with acetaminophen (for example, 25-50 mg diphenhydramine and 500-650 mg acetaminophen) within approximately 30 to 60 minutes prior to dosing of M7824 is optional and at the discretion of the Investigator.

#### 3.2.3 NHS-IL12

NHS-IL12 will be administered at as dose of 16.8mcg/kg by SC injection every 4 weeks for up to 4 consecutive doses then 8mcg/kg every 4 weeks thereafter. However lower doses may also be used as per Section 3.4.3. The dose of NHS-IL12 will be calculated based on the weight of the


subject determined within 2 weeks prior to the day of drug administration. The dose of NHS-IL12 used for the previous administration can be repeated if the change in the subject's weight is 10% or less than the weight used for the last dose calculation.

#### 3.3 STUDY INTERVENTION COMPLIANCE

All study interventions will be given at NIH and documented in the electronic medical record.

#### 3.4 DOSE MODIFICATIONS

#### 3.4.1 Discontinuation

Treatment with individual agents will be discontinued in the case of:

- Any Grade 4 or higher adverse drug reactions (ADRs) as defined by CTCAE v5.0 and assessed as possibly related to that agent by the Investigator, except for laboratory values that are asymptomatic or resolve to Grade ≤ 1 or baseline grade within 7 days
- Any Grade 3 ADRs possibly attributed to an agent except for any of the following:
  - Grade 3 flu-like symptoms or fever, as well as associated symptoms of fatigue, headaches, nausea, emesis which can be controlled with conservative medical management.
  - o Tumor flare phenomenon defined as local pain, irritation, or rash localized at sites of known or suspected tumor.
  - o Grade 3 Hgb decrease (< 8.0 g/dL) that is clinically manageable with blood transfusions or erythroid growth factor use does not require treatment discontinuation.
  - o Grade 3 laboratory values that are asymptomatic or resolve to Grade  $\leq 1$  or baseline grade within 14 days.
  - o Keratoacanthoma and squamous cell carcinoma of the skin.
  - o Any endocrinopathy that can be medically managed with hormone replacement
  - o Any grade 3 adverse drug reaction which can be medically managed with minimal risk to the participant (e.g., placement of a pleural catheter for recurrent inflammatory pleural effusions) and resolves to at least grade one or baseline grade within 14 days.

#### 3.4.2 Dose Delay

Individual agents should be withheld for any Grade 2 or 3 ADR possibly attributed to that agent until resolution to Grade  $\leq 1$  unless the ADR in the opinion of the investigator is not clinically relevant or can be medically managed with minimal risk to the participant. NHS-IL12 may be restarted at any scheduled visit as long as there is at least 11 days between doses of this agent. Should a clinically relevant grade 2 or 3 ADR persist for more than 4 weeks, consideration should be given to discontinuing treatment with that individual agent at the discretion of the investigator.

For non-medical logistical reasons, unrelated acute illnesses, or palliative radiation, scheduled assessments and dosing can be delayed up to 2 months. Where at all possible, dosing should be restarted to keep in line with the original treatment schedule.

#### 3.4.3 Dose Modification

Participants with dose modifications or skipped doses within DLT period for reasons other than a DLT (e.g., logistical reasons) who do not experience a DLT within the DLT window will not be evaluable for DLTs and will be replaced for the six-participant lead in DLT assessment.


Participants who have dose modifications or skipped doses within the DLT period for logistical reasons and nevertheless experience a DLT within the DLT period will be considered DLT evaluable.

PDS0101 HPV vaccine: Vaccine doses will not be modified but doses may be skipped per investigator discretion. For example, PDS0101 (which targets HPV 16 specifically) may be held for non-HPV 16 tumors per investigator discretion.

M7824: Doses (including starting doses) may be reduced to a 300 or 600 mg flat dose or doses may be skipped.

NHS-IL12: All patients, except patients with cervical cancer and prior pelvic radiation and brachytherapy (described in the next paragraph), will receive NHS-IL12 at a starting dose of 16.8 mcg/kg for up to a total of 4 consecutive doses at which time the dose will be reduced to 8 mcg/kg thereafter. Doses may be reduced to 8 mcg/kg at any time after the first dose for grade ≥ 2 flu-like symptoms, fever, or other NHS-IL12 related toxicities. Additionally, doses may be skipped or further dose-reduced to 4 or 6 mcg/kg. For patients who have already received initial starting doses of NHS-IL12 at 8 mcg/kg they may receive NHS-IL12 at 16.8 mcg/kg for up to a total of 4 consecutive doses. In select participants receiving doses of 8 mcg/kg or lower, consideration may be given to every 2 week dosing of this agent.

In patients with cervical cancer with prior pelvic radiation and boost brachytherapy where a potential higher risk of grade 3 hematuria may exist with the full starting doses of M7824 at 1200 mg and NHS-IL12 at 16.8 mcg/kg, a staring dose of M7824 at 600 mg and NHS-IL12 at 4 mcg/kg will be used instead. If grade 3 or greater hematuria occurs in  $\geq$  2 out of four of these patients then the starting dose for these patients will be lowered to M7824 at 300 mg and NHS-IL12 at 4 mcg/kg. If grade 3 or greater hematuria occurs in  $\geq$  2 out of four of these patients when given M7824 at 300 mg and NHS-IL12 at 4 mcg/kg then these patients will no longer to be eligible to enroll on this protocol. On the other hand, if  $\leq$  2 patients out of four have grade 3 or greater bleeding events when given M7824 at 600 mg and NHS-IL12 at 4 mcg/kg but objective responses are also observed in  $\leq$  2 out of these four patients then a dose of M7824 at 1200 mg in combination with NHS-IL12 at 4 mcg/kg will be evaluated in these patients. If  $\geq$  2 patients out of four have grade 3 or greater bleeding events or  $\leq$  2 out of four patients have objective responses when given M7824 at 1200 mg and NHS-IL12 at 4 mcg/kg then the combination of M7824 at 600 mg and NHS-IL12 at 6 mcg/kg may be evaluated.

Stopping Rule: If more than one third of enrolled patients have permanently discontinued one or more study agents due to grade 3 or 4 toxicity per guidelines in Section 3.4.1 or any death has occurred which is at least possibly related to study regimen this will prompt a suspension of accrual and reassessment of available safety information prior to reopening study to accrual.


# 3.4.4 Guidelines for Management of Infusion Reactions

| NCI-CTCAE Grade | Treatment Modification for Infused Agent (M7824) |
|---|---|
| Grade 1 – mild Mild transient reaction; infusion interruption not indicated; intervention not indicated. | Consider decreasing the infusion rate of the particular agent by 50% and monitoring closely for any worsening. |
| Grade 2 – moderate Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDs, narcotics, i.v. fluids); prophylactic medications indicated for ≤ 24 hours. | Consider temporarily discontinuing infusion of the particular agent. Consider resuming infusion of the particular agent at 50% of previous rate once infusion related reaction has resolved or decreased to at least Grade 1 in severity, and monitor closely for any worsening. |
| Grade 3 or Grade 4 – severe or life-threatening Grade 3: Prolonged (e.g., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); hospitalization indicated for clinical sequelae. Grade 4: Life-threatening consequences; urgent intervention indicated. | Stop the infusion immediately and disconnect infusion tubing from the subject. For grade 3 events: Consider withdrawing immediately from treatment with that particular agent and not offering any further treatment with that agent based upon if the clinical condition can be safely managed. For grade 4 events: Withdraw immediately from treatment and do not offer further treatment with that agent. |

If the infusion rate of M7824 has been decreased by 50% or interrupted due to an infusion reaction, keep it decreased for the next scheduled infusion. If no infusion reaction is observed in the next scheduled infusion, the infusion rate may be returned to baseline at the subsequent infusions based on investigator's medical judgment.

If hypersensitivity reaction occurs, the subject should be treated according to the best available medical practice.

# 3.4.5 Guidelines for Management of Immune-Mediated Adverse Reactions

(In addition to the below guidelines, investigators may also use NCCN, ASCO, SITC or FDA guidelines for Immune Related Adverse Events)

| | Gastrointestinal irAEs | |
|---|---|---|
| Severity of Diarrhea/Colitis<br>(NCI-CTCAE v5) | Initial Management | Follow-up Management |
| Grade 1 Diarrhea: < 4 stools/day over Baseline Colitis: asymptomatic | Consider continuing M7824 Symptomatic treatment (e.g. loperamide) | Consider close monitoring for worsening symptoms Consider educating subject to report worsening immediately If worsens: Treat as Grade 2, 3 or 4. |
| Grade 2 Diarrhea: 4 to 6 stools per day over Baseline; IV fluids indicated < 24 hours; not interfering with ADL Colitis: abdominal pain; blood in stool | Consider withholding M7824 Symptomatic treatment | If improves to Grade ≤ 1: Consider resuming therapy If persists > 7 days or recurs: Consider treating as Grade 3 or 4. |
| Grade 3 to 4 Diarrhea (Grade 3): ≥ 7 stools per day over Baseline; incontinence; IV fluids ≥ 24 h; interfering with ADL Colitis (Grade 3): severe abdominal pain, medical intervention indicated, peritoneal signs Grade 4: life-threatening, perforation | Consider withholding or permanently discontinuing M7824 for Grade 3 events based upon if the clinical condition can be safely managed. For grade 4 events permanently discontinue treatment. Consider 1.0 to 2.0 mg/kg/day prednisone IV or equivalent Consider adding prophylactic antibiotics for opportunistic infections Consider lower endoscopy | If improves: Consider continuing steroids until Grade ≤ 1, then tapering over at least 1 month; consider resuming therapy following steroids taper (for initial Grade 3). If worsens, persists > 7 days, or recurs after improvement: Consider adding infliximab 5mg/kg (if no contraindication). Note: infliximab should not be used in cases of perforation or sepsis. |

| Dermatological irAEs | | |
|---|---|---|
| Grade of Rash<br>(NCI-CTCAE v5) | Initial Management | Follow-up Management |
| Grade 1 to 2 Covering ≤ 30% body surface area | Consider continuing M7824 Consider symptomatic therapy (for example, antihistamines, topical steroids) | If persists > 1 to 2 weeks or recurs: Consider withholding M7824 therapy Consider skin biopsy |
| | | Consider 0.5-1.0 mg/kg/day prednisone or equivalent. Once improving, consider tapering steroids over at least 1 month, consider prophylactic antibiotics for opportunistic infections, and consider resuming M7824 therapy following steroids taper. If worsens: Consider treating as Grade 3 to 4. |
| Grade 3 to 4 Grade 3: Covering > 30% body surface area; Grade 4: Life threatening consequences | Consider withholding or permanently discontinuing M7824 for Grade 3 events based upon if the clinical condition can be safely managed. For grade 4 events permanently discontinue treatment. Consider skin biopsy Consider dermatology consult Consider 1.0 to 2.0 mg/kg/day prednisone or equivalent Consider adding prophylactic | If improves to Grade ≤ 1:<br>Consider tapering steroids over at<br>least 1 month; consider resuming<br>therapy following steroids taper<br>(for initial Grade 3). |
| | antibiotics for opportunistic infections | |
| | Pulmonary irAEs | |
| Grade of Pneumonitis<br>(NCI-CTCAE v5) | Initial Management | Follow-up Management |
| Grade 1 Radiographic changes only | Consider withholding M7824<br>Consider Pulmonary and Infectious<br>Disease consults | Consider re-assessing at least every 3 weeks If worsens: Consider treating as Grade 2 or Grade 3 to 4. |
| Grade 2 Mild to moderate new symptoms | Consider withholding M7824 | If improves: |

| Crade of Liver Test Flavation | Hepatic irAEs | |
|---|---|---|
| Grade 3 to 4 Grade 3: Severe new symptoms; New/worsening hypoxia; Grade 4: Life-threatening | Consider withholding or permanently discontinuing M7824 for Grade 3 events based upon if the clinical condition can be safely managed. For grade 4 events permanently discontinue treatment. Consider hospitalization. Consider pulmonary and Infectious Disease consults. Consider 1.0 to 2.0 mg/kg/day prednisone or equivalent Consider adding prophylactic antibiotics for opportunistic infections Consider bronchoscopy, lung biopsy | If improves to Grade ≤ 1: Consider tapering steroids over at least 1 month If not improving after 48 hours or worsening: Consider adding additional immunosuppression (for example, infliximab, cyclophosphamide, IV immunoglobulin, or mycophenolate mofetil) |
| | Consider pulmonary and Infectious Disease consults Consider monitoring symptoms daily; consider hospitalization Consider 1.0 to 2.0 mg/kg/day prednisone or equivalent Consider adding prophylactic antibiotics for opportunistic infections Consider bronchoscopy, lung biopsy | When symptoms return to Grade ≤ 1, consider tapering steroids over at least 1 month, and then consider resuming therapy following steroids taper If not improving after 2 weeks or worsening: Consider treating as Grade 3 to 4. |

| Grade of Liver Test Elevation<br>(NCI-CTCAE v5) | Initial Management | Follow-up Management |
|---|---|---|
| Grade 1 Grade 1 AST or ALT > ULN to 3.0 x ULN and/or Total bilirubin > ULN to 1.5 x ULN | Consider continuing M7824 | Consider continued liver function monitoring If worsens: Consider treating as Grade 2 or 3 to 4. |
| Grade 2 AST or ALT > 3.0 to $\leq$ 5 x ULN and/or total bilirubin > 1.5 to $\leq$ 3 x ULN | Consider withholding M7824 | If returns to Grade ≤ 1: Consider resuming therapy. If elevation persists > 7 days or worsens: Consider treating as Grade 3 to 4. |
| Grade 3 to 4 AST or ALT > 5 x ULN and/or total bilirubin > 3 x ULN | Consider withholding or permanently discontinuing M7824 for Grade 3 events based upon if the clinical condition can be safely managed. For grade 4 events permanently discontinue treatment. | If returns to Grade ≤ 1:<br>Consider tapering steroids over at<br>least 1 month<br>If does not improve in > 7 days,<br>worsens or rebounds: |

| | Consider 1.0 to 2.0 mg/kg/day prednisone or equivalent Consider adding prophylactic antibiotics for opportunistic infections Consider consulting gastroenterologist/ hepatologist Consider obtaining MRI/CT scan of liver and liver biopsy if clinically warranted | Consider adding mycophenolate mofetil 1 gram (g) twice daily If no response within an additional 7 days, consider other immunosuppressants per local guidelines. |
|---|---|---|
| | Renal irAEs | |
| Grade of Creatinine Increased<br>(NCI-CTCAE v5) | Initial Management | Follow-up Management |
| Grade 1 Creatinine increased > ULN to 1.5 x ULN | Consider continuing M7824 | Continue renal function monitoring If worsens: Consider treating as Grade 2 to 3 or 4. |
| Grade 2 Creatinine increased > 1.5 and $\leq 6 \text{ x}$ ULN | Consider withholding M7824 Consider 1.0 to 2.0 mg/kg/day prednisone or equivalent. Consider adding prophylactic antibiotics for opportunistic infections Consider renal biopsy | If returns to Grade ≤1: Consider tapering steroids over at least 1 month, and consider resuming therapy following steroids taper. If worsens: Treat as Grade 4. |
| Grade 3-4 Creatinine increased > 6 x ULN | Consider withholding or permanently discontinuing M7824 for Grade 3 events based upon if the clinical condition can be safely managed. For grade 4 events permanently discontinue treatment. Consider 1.0 to 2.0 mg/kg/day prednisone or equivalent. Consider adding prophylactic antibiotics for opportunistic infections Consider renal biopsy Consider Nephrology consult | If returns to Grade ≤1: Consider tapering steroids over at least 1 month. |


| Cardiac irAEs | | |
|---|---|---|
| Myocarditis | Myocarditis Initial Management Follow-up Managem | |
| New onset of cardiac signs or symptoms and / or new laboratory cardiac biomarker elevations (e.g. troponin, CK-MB, BNP) or cardiac imaging abnormalities suggestive of myocarditis. | Consider withholding or permanently discontinuing M7824 based upon if the clinical condition can be safely managed. Consider hospitalization In the presence of life threatening cardiac decompensation, consider transfer to a facility experienced in advanced heart failure and arrhythmia management. Consider cardiology consult to establish etiology and rule-out immune-mediated myocarditis. Consider myocardial biopsy if recommended per cardiology consult. | If symptoms improve and immune-mediated etiology is ruled out, consider re-starting therapy. If symptoms do not improve/worsen, viral myocarditis is excluded, and immune-mediated etiology is suspected or confirmed following cardiology consult, consider managing as immune-mediated myocarditis. |
| Immune-mediated myocarditis | Consider withholding or permanently discontinuing M7824 based upon if the clinical condition can be safely managed. Consider guideline based supportive treatment as appropriate as per cardiology consult. Consider 1.0 to 2.0 mg/kg/day prednisone or equivalent Consider adding prophylactic antibiotics for opportunistic infections. | Once improving, consider tapering steroids over at least 1 month. If no improvement or worsening, consider additional immunosuppressants (e.g. azathioprine, cyclosporine A). |

<sup>\*</sup>Local guidelines, or eg. ESC or AHA guidelines

ESC guidelines website: https://www.escardio.org/Guidelines/Clinical-Practice-Guidelines

AHA guidelines website:

http://professional.heart.org/professional/GuidelinesStatements/searchresults.jsp?q=&y=&t=1001

| Endocrine ir AEs | | |
|---|---|---|
| Endocrine Disorder Initial Management Follow-up Management | | |
| Grade 1 or Grade 2<br>endocrinopathies (hypothyroidism,<br>hyperthyroidism, adrenal<br>insufficiency, type I diabetes<br>mellitus) | Consider continuing M7824 Consider endocrinology consult if needed | Consider continuing hormone replacement/suppression and monitoring of endocrine function as appropriate. |

| Grade 3 or Grade 4 endocrinopathies (hypothyroidism, hyperthyroidism, adrenal insufficiency, type I diabetes mellitus) | Consider starting thyroid hormone replacement therapy (for hypothyroidism), anti-thyroid treatment (for hyperthyroidism), corticosteroids (for adrenal insufficiency) or insulin (for Type I diabetes mellitus) as appropriate. Consider ruling-out secondary endocrinopathies (i.e. hypopituitarism / hypophysitis) Consider withholding or permanently discontinuing M7824 for Grade 3-4 events based upon if the clinical condition can be safely managed. Consider hospitalization Consider endocrinology consult Consider starting thyroid hormone replacement therapy (for hypothyroidism), anti-thyroid treatment (for hyperthyroidism), corticosteroids (for adrenal insufficiency) or insulin (for type I diabetes mellitus) as appropriate. | Consider resuming therapy once symptoms and/or laboratory tests improve to Grade ≤ 1 (with or without hormone replacement/suppression). Consider continuing hormone replacement/suppression and monitoring of endocrine function as appropriate. |
|---|---|---|
| Hypopituitarism/Hypophysitis (secondary endocrinopathies) | Consider ruling-out secondary endocrinopathies (i.e. hypopituitarism / hypophysitis) If secondary thyroid and/or adrenal insufficiency is confirmed (i.e. subnormal serum FT4 with inappropriately low TSH and/or low serum cortisol with inappropriately low ACTH): Consider referring to endocrinologist for dynamic testing as indicated and measurement of other hormones (FSH, LH, GH/IGF-1, PRL, testosterone in men, estrogens in women) Consider hormone replacement/suppressive therapy as appropriate Consider performing pituitary MRI and visual field examination as indicated If hypophysitis confirmed: | Consider resuming therapy once symptoms and hormone tests improve to Grade ≤ 1 (with or without hormone replacement). In addition, for hypophysitis with abnormal MRI, consider resuming M7824 only once shrinkage of the pituitary gland on MRI/CT scan is documented. Consider continuing hormone replacement/suppression therapy as appropriate. |

| | <ul> <li>Continue M7824 if mild symptoms</li> <li>Consider withholding M7824 and if moderate, severe or lifethreatening symptoms of hypophysitis. Consider hospitalization. Consider initiating corticosteroids (1 to 2 mg/kg/day prednisone or equivalent) followed by corticosteroids taper during at least 1 month.</li> <li>Consider adding prophylactic antibiotics for opportunistic infections.</li> </ul> | |
|---|---|---|
| | Other irAEs (not described above) | |
| Grade of other irAEs<br>(NCI-CTCAE v5) | Initial Management | Follow-up Management |
| Grade 2 or Grade 3 clinical signs or symptoms suggestive of a potential irAE | Consider withholding M7824 pending clinical investigation | If irAE is ruled out, consider managing as appropriate according to the diagnosis and consider re-starting therapy If irAE is confirmed, consider treating as Grade 2 or 3 irAE. |
| Grade 2 irAE or first occurrence of Grade 3 irAE | Consider withholding M7824 based upon if the clinical condition can be safely managed. Consider 1.0 to 2.0 mg/kg/day prednisone or equivalent Consider adding prophylactic antibiotics for opportunistic infections Specialty consult as appropriate | If improves to Grade ≤ 1: Consider tapering steroids over at least 1 month and resuming therapy following steroids taper. |
| Recurrence of same Grade 3 irAEs | Consider permanently discontinuing M7824 based upon if the clinical condition can be safely managed; Consider 1.0 to 2.0 mg/kg/day prednisone or equivalent Consider adding prophylactic antibiotics for opportunistic infections Specialty consult as appropriate | If improves to Grade ≤ 1: Consider tapering steroids over at least 1 month. |


| Grade 4 | Permanently discontinue M7824 Consider to 2.0 mg/kg/day prednisone or equivalent and/or other immunosuppressant as needed Consider adding prophylactic antibiotics for opportunistic infections Consider specialty consult as appropriate | If improves to Grade ≤ 1:<br>Consider tapering steroids over<br>at least 1 month |
|---|---|---|
| Requirement for 10 mg per day or greater prednisone or equivalent for more than 12 weeks for reasons other than hormonal replacement for adrenal insufficiency Persistent Grade 2 or 3 irAE | Consider permanently discontinuing M7824 Consider specialty consult as appropriate | |
| lasting 12 weeks or longer | | |

Abbreviations: ACTH=adrenocorticotropic hormone; ADL=activities of daily living; ALT=alanine aminotransferase; AST=aspartate aminotransferase; BNP=B-type natriuretic peptide; CK-MB=creatine kinase MB; CT= computed tomography; FSH=follicle-stimulating hormone; GH=growth hormone; IGF-1=insulin-like growth factor 1; irAE=immune related adverse event; IV=intravenous; LH=luteinizing hormone; MRI=magnetic resonance imaging; NCI CTCAE=National Cancer Institute Common Terminology Criteria for Adverse Events; PRL=prolactin; T4=thyroxine; TSH=thyroid stimulating hormone; ULN=upper limit of normal


# 3.5 STUDY CALENDAR

| Procedure | Screening <sup>1</sup> | Baseline /<br>Week 1 <sup>2</sup> | Week (2N+1) <sup>3</sup> | EOT <sup>4</sup> | Safety<br>follow<br>up <sup>5</sup> | Long<br>Term<br>follow up <sup>6</sup> |
|---|---|---|---|---|---|---|
| Treatment <sup>3</sup> | | X | X | | | |
| NIH Advance Directives Form <sup>7</sup> | | X | | | | |
| Medical History | X | | | | | |
| Height | X | | | | | |
| Physical exam, weight, vital signs, ECOG | X | X | X | X | X | |
| HIV, HCV, HepB | X | | | | | |
| EKG | X | | | X | X | |
| CBC with differential | X | X | X | X | X | |
| Biochemical profile <sup>8</sup> | X | X | X | X | X | |
| Tumor Markers <sup>9</sup> | | X | X | X | | |
| CD4 <sup>10</sup> | X | | | | | |
| HLA typing | X | | | | | |
| ACTH, TSH, reflex Free T4, lipase, amylase, CRP | | X | X <sup>11</sup> | | | |
| Urinalysis | X | | | | | |
| Urine or serum pregnancy<br>testing in women of<br>childbearing potential | X | X | X | | | |
| PT, INR, aPTT | | X | | | | |
| Tumor evaluation (CT Scan) <sup>12</sup> | X | | X | | | X |
| Brain CT <sup>13</sup> | X | | | | | |
| Concomitant Medications | | X | X | X | X | |
| Adverse events | | X | X | X | X | |
| Optional biopsy for immune analysis <sup>14</sup> | | X | X | | | |
| Research Blood 15 | | X | X | X | | |
| Telephone Follow Up | | | | | X | X |


1. Screening evaluations performed within 28 days prior to the first drug administration, unless specified in Section 2.2.

- 2. Baseline evaluations performed within 1 week prior to first drug administration.
- 3. Schedule of therapeutic agents administered will be as outlined in Section 3.1, Figure 19.. NHS-IL12 will be given every 4 weeks, M7824 infusion will be every two weeks and HPV vaccine will be given every 4 weeks for the first 6 doses followed by every 12 weeks thereafter. (The first administration of HPV vaccine should preferably be given 1-2 weeks before the first administration of NHS-IL12 and M7824.) Administration of study agents and indicated evaluations can be done up to 14 days earlier or delayed up to 14 days due to holidays, inclement weather, conflicts, or similar reasons. The timing of subsequent administrations is adjusted to maintain a minimum of 11 days between treatments of similar agents.
- 4. EOT End of treatment visit: Where feasible, on the day of or within 7 days of the decision to discontinue treatment prematurely before completion of one year of treatment. Does not need to be completed if drug is withheld after one year of treatment.
- 5. 28 days (+/- 7 days) after last treatment. If subjects are not willing to come to NIH to FU visit, they will be contacted by phone to assess adverse events.
- 6. Participants who have come off treatment for disease progression will be followed by phone annually for survival. Participants who have not progressed on treatment will continue to be followed and scanned per investigator discretion until progression. Those that completed one year of treatment will be invited for an additional year of treatment at the time of progression. Initial and follow up courses of treatment may extend beyond a year per investigator discretion.
- 7. As indicated in Section 12.3, all subjects will be offered the opportunity to complete an NIH advanced directives form. This should be done preferably at baseline but can be done at any time during the study as long as the capacity to do so is retained. The completion of the form is strongly recommended, but is not required.
- 8. Biochemical profile: mineral panel, sodium, potassium, chloride, bicarbonate, calcium, glucose, BUN, creatinine, ALT, AST, alkaline phosphatase, total protein, albumin, and total and direct bilirubin. Note: the mineral panel will start from baseline onward.
- 9. Evaluate CEA, CA19-9, CA125 and CA15-3 at baseline and follow elevated values thereafter.
- 10. In HIV positive participants.
- 11. Every 8 weeks.
- 12. Every 8 weeks. In the event of a PR or CR tumor imaging assessments may be performed every 3 months (+/- 2 weeks) at the discretion of the investigator. Tumor assessment should be continued beyond end of treatment in participants who have not experience PD until they experience PD in order to assess PFS. MRI will be used when CT scan is not an option to follow the disease clinically. Gadolinium will be used only for clinically indicated MRIs. Bone scans and other imaging assessments may also be performed as clinically indicated.
- 13. In participants with known CNS disease as described in Section 2.1.2.4. MRIs may be performed as clinically indicated in this population.
- 14. Optional biopsies at baseline and as close as possible to first imaging restaging.
- 15. Where feasible, research blood for study assessments (see Section 5) will be collected at baseline, 3 days and 1 week after the first M7824 + NHS-IL12 dose) as well as at weeks 3 and 7 and at restaging visits in selected participants, per PI discretion.


#### 3.6 COST AND COMPENSATION

#### 3.6.1 Costs

NIH does not bill health insurance companies or participants for any research or related clinical care that participants receive at the NIH Clinical Center. If some tests and procedures are performed outside the NIH Clinical Center, participants may have to pay for these costs if they are not covered by an insurance company. Medicines that are not part of the study treatment will not be provided or paid for by the NIH Clinical Center.

### 3.6.2 Compensation

There will be no compensation provided on this study.

#### 3.6.3 Reimbursement

The NCI will cover the costs of some expenses associated with protocol participation. Some of these costs may be paid directly by the NIH and some may be reimbursed to the participant/guardian as appropriate. The amount and form of these payments are determined by the NCI Travel and Lodging Reimbursement Policy.

# 3.7 CRITERIA FOR REMOVAL FROM PROTOCOL THERAPY AND OFF STUDY CRITERIA

Regardless of reason for removal from study therapy, participants will be asked to have a 28 day follow up safety visit. Participants who refuse to return for this visit will be asked to review any safety concerns by phone within this time period.

# 3.7.1 Criteria for Removal from Protocol Therapy

- Clinical or radiographic progression of disease except when the investigator feels the subject is still benefiting from treatment. (It is generally preferable for participants to remain on treatment past initial radiographic progression in case there is pseudo progression, except when the investigator feels that the clinical picture warrants changing therapy at initial progression).
- Unacceptable Toxicity possibly attributed to all active therapies.
- Participant requests to be withdrawn from active therapy.
- Start of another systemic anticancer treatment or participation in another investigational therapeutic trial. Focal palliative radiotherapy, ablation, or surgery to a site of disease will not necessitate removal from protocol therapy.
- Investigator discretion.
- Positive pregnancy test.

# 3.7.2 Off-Study Criteria

- Screen failure.
- PI decision to end the study.
- Participant requests to be withdrawn from study.
- Participant lost to follow up.


- Investigator discretion.
- Death.

## 3.7.3 Lost to Follow-up

A participant will be considered lost to follow-up if he or she fails to return for 4 scheduled visits and is unable to be contacted by the study site staff.

The following actions must be taken if a participant fails to return to the clinic for a required study visit:

- The site will attempt to contact the participant and reschedule the missed visit for within the next 2 weeks and counsel the participant on the importance of maintaining the assigned visit schedule and ascertain if the participant wishes to and/or should continue in the study.
- Before a participant is deemed lost to follow-up, the investigator or designee will make
  every effort to regain contact with the participant (where possible, 3 telephone calls and, if
  necessary, an IRB approved certified letter to the participant's last known mailing address
  or local equivalent methods). These contact attempts should be documented in the
  participant's medical record or study file.
- Should the participant continue to be unreachable, he or she will be considered to have withdrawn from the study with a primary reason of lost to follow-up.

#### 4 CONCOMITANT MEDICATIONS/MEASURES

Any medications (other than those excluded by the clinical trial protocol) that are considered necessary to protect subject welfare or alleviate symptoms and will not interfere with the trial medication may be given at the Investigator's discretion.

Palliative radiotherapy delivered in a normal organ-spearing technique may be administered during the trial. The assessment of PD will not be based on the necessity for palliative radiotherapy.

#### 4.1 THE FOLLOWING TREATMENTS SHOULD NOT BE ADMINISTERED DURING THE TRIAL

- Other immunotherapies or immunosuppressive drugs (for example, chemotherapy or systemic corticosteroids except for prophylaxis or treatment of allergic reactions, endocrine replacement therapy at low dose prednisone [≤ 10 mg daily] or equivalent, for the treatment of irAEs, or for short courses (≤ 14 days) as appropriate medical therapy for unrelated medical conditions (e.g., asthma). Steroids with no or minimal systemic effect (topical, inhalation) are allowed.
- Prophylactic use of corticosteroids for infusion related reactions. Corticosteroid administration prior to CT scans in participants with intravenous contrast allergy is allowed.
- Any live vaccine therapies for the prevention of infectious disease. Administration of
  inactivated vaccines is allowed (for example, inactivated influenza vaccines or locally
  approved COVID vaccines).
- Systemic anticancer treatment.


# 5 CORRELATIVE STUDIES FOR RESEARCH/PHARMACOKINETIC STUDIES

# 5.1 BIOSPECIMEN COLLECTION

| Test/assay | Volume<br>(approx.) per<br>Timepoint | Type of tube <sup>a</sup> | Collection point | Location of specimen analysis* |
|---|---|---|---|---|
| Standard and 123 immune cell subsets by FACS | | | See study calendar 3.5 | LTIB |
| Functional<br>Analysis of<br>immune cell<br>subsets by FACS | 60-80 mL<br>blood for<br>PBMCs | Sodium heparin (green top) tubes | | LTIB |
| Antigen Specific<br>Immune Response<br>by cytokine<br>staining assay | | | | LTIB |
| T cell clonality by immunseq platform | | | | LTIB and NCI<br>Frederick<br>Genomic Core<br>Facility |
| RNA expression level of 770 genes | | | | LTIB and NCI<br>Frederick<br>Genomic Core<br>Facility |
| Soluble Factors<br>(to include sCD27<br>and sCD40<br>ligand) by ELISA | 16 mL blood<br>for serum | SST | | LTIB |
| Immune Markers by IHC | Tumor samples | N/A | | GMB TIME Lab |
| RNA expression level of 770 genes | Tumor samples | N/A | | LTIB and NCI<br>Frederick<br>Genomic Core<br>Facility |


| Test/assay | Volume<br>(approx.) per<br>Timepoint | Type of tube <sup>a</sup> | Collection point | Location of specimen analysis* |
|---|---|---|---|---|
| HPV status by PCR of DNA | Tumor samples | N/A | | Dr. Hinrich's Lab |
| Circulating tumor<br>DNA (ctDNA) by<br>PCR system | Plasma | EDTA (lavender top) | | LTIB and NIH<br>Core Facility |
| T cell clonality by immunoseq platform | Tumor<br>samples | N/A | | LTIB and NCI<br>Frederick<br>Genomic Core<br>Facility |

<sup>&</sup>lt;sup>a</sup> Please note that tubes and media may be substituted based on availability with the permission of the PI or laboratory investigator.

## 5.1.1 Immune Phenotyping

Exploratory immunologic studies will be conducted to evaluate the study drug's effect on the immune response before and after treatment, to gain insight into potential biomarkers, and help improve the administered therapy. Blood will be collected as per Study Calendar 3.5. The following immune assays may be performed at the Laboratory of Tumor Immunology and Biology (LTIB) at the NCI's Center for Cancer Research (CCR) in select participants where adequate samples are available:

- 1. PBMCs may be analyzed for changes in standard immune cell types (CD4 and CD8 T cells, natural killer [NK] cells, regulatory T cells [Tregs], myeloid-derived suppressor cells [MDSCs], and dendritic cells) as well as 123 immune cell subsets, using multi-color flow cytometry.
- 2. PBMCs from selected subjects may be analyzed for function of specific immune cell subsets, including CD4 and CD8 T cells, NK cells, Tregs, and MDSCs using flow-based assays.
- 3. PBMCs may be analyzed for tumor antigen-specific immune responses using an intracellular cytokine staining assay. PBMCs will be stimulated in vitro with overlapping 15-mer peptide pools encoding the tumor-associated antigens such as CEA, MUC-1 and Brachyury; control peptide pools will involve the use of human leukocyte antigen peptide as a negative control and CEFT peptide mix as a positive control. CEFT is a mixture of peptides of CMV, Epstein-Barr virus, influenza, and tetanus toxin. Post-stimulation analyses of CD4 and CD8 T cells will involve the production of IFN-γ, IL-2, TNF, and the degranulation marker CD107a. If sufficient PBMCs are available, assays may also be performed for the development of T cells to other tumor-associated antigens.

<sup>\*</sup>Research blood samples will be sent to the Clinical Services Program – Leidos Biomedical Research, Inc. (CSP) (Section 5.3.1) for barcoding, initial processing and storage. Tissue will be sent to the Laboratory of Pathology as described in Section 5.3.2. From these facilities, coded, linked samples will be sent to the designated labs for analysis upon request.


#### 5.1.2 Soluble Factors

Samples for soluble factor analysis will be collected as per Study Calendar 3.5.

-Sera may be analyzed pre- and post-therapy for the following soluble factors: sCD27, sCD40 ligand using commercial ELISA kits.

-Sera may be analyzed for changes in cytokines (IFN-γ, IL-10, IL-12, IL-2, IL-4, etc.), chemokines, antibodies, tumor-associated antigens, and/or other markers using ELISA or multiplexed assays (e.g., Mesoscale, Luminex, cytokine bead array).

## 5.1.3 Analyses of Tumor Tissue for Immune Markers

Study of immune infiltration as well as PD-L1 status within the tumor microenvironment pre vs. post treatment by IHC and/or multiplex immunofluorescence may be performed by the GMB TIME Lab. Where available, archival tumor samples will be requested (preferably tissue samples from the last 6 months). For participants with lesions amenable to biopsy, two optional biopsies may be performed at baseline and at first restaging. Tumor samples will be sent to the Laboratory of Pathology for disease evaluation; remaining samples will be used for research. Tissue samples for research may also be stored in CSP as described in Section **5.3.1**.

#### 5.1.4 Assessment of HPV status

In participants with available tumor tissue (either archival or by optional biopsy), HPV testing will be performed using the Roche Cobas or Becton Dickinson HPV PCR based DNA assay, if no prior HPV testing of the tumor has been performed. This will be done through collaboration with Dr. Hinrich's Lab.

# 5.1.5 Circulating tumor DNA

If sufficient plasma is available, selected participant samples may be analyzed for circulating tumor DNA (LTIB and NIH Core Facility). Plasma DNA will be isolated with an automated purification system by Promega Corp using a system-attached bar-code reader to track samples and DNA products. The circulating tumor/HPV DNA will be quantified with a digital droplet PCR system from Bio-Rad to obtain precise quantification. This is just quantification by PCR. There is no DNA sequencing.

#### 5.2 SAMPLES FOR GENETIC/GENOMIC ANALYSIS

# 5.2.1 Description of the scope of genetic/genomic analysis

#### 5.2.1.1 RNA and T-cell Receptor Clonality Analysis of Blood and Tumor Tissue

Where possible, RNA expression and T-cell receptor clonality analysis will be done on the peripheral blood as well as archived tumor tissue or optional biopsies to help further evaluate changes in immune response and RNA expression levels with treatment as well as to determine tumor and infiltrating lymphocyte characteristics which may be predictive of response to treatment. In addition, these analyses will also be used to gauge resistance mechanisms and additional targets for future therapy. Coded, linked samples may be analyzed for RNA expression levels using the Nanostring platform and T-cell receptor clonality using the ImmunoSeq platform (LTIB and NCI Frederick Genomic Core Facility).

NCI Fredrick Genomic Core Facility:


Leidos Biomedical Research, Inc:

Dr. Xiaolin Wu ATRF, Rm C3016 8560 Progress Drive Frederick, MD 21701 Ph. 301-846-7677

5.2.2 Description of how privacy and confidentiality of medical information/biological specimens will be maximized

Confidentiality for genetic samples will be maintained as described (Section 5.3.1 and 5.3.2).

# 5.2.3 Management of Results

Subjects will be contacted if a clinically actionable gene variant is discovered. Clinically actionable findings for the purpose of this study are defined as disorders appearing in the American College of Medical Genetics and Genomics recommendations for the return of incidental findings that is current at the time of primary analysis. (A list of current guidelines is maintained on the CCR intranet: <a href="https://ccrod.cancer.gov/confluence/display/CCRCRO/Incidental+Findings+Lists">https://ccrod.cancer.gov/confluence/display/CCRCRO/Incidental+Findings+Lists</a>). Subjects will be contacted at this time with a request to provide a blood sample to be sent to a CLIA certified laboratory. If the research findings are verified in the CLIA certified lab, the subject will be offered the opportunity to come to NIH (at our expense) to have genetic education and counseling to explain this result. If the subject does not want to come to NIH, a referral to a local genetic healthcare provider will be provided (at their expense).

This is the only time during the course of the study that incidental findings will be returned. No interrogations regarding clinically actionable findings will be made after the primary analysis.

#### 5.3 SAMPLE STORAGE, TRACKING AND DISPOSITION

Samples will be ordered in CRIS and tracked through a Clinical Trial Data Management system. Should a CRIS screen not be available, the CRIS downtime procedures will be followed. Samples will not be sent outside the National Institutes for Health (NIH) appropriate approvals and/or agreements, if required.

5.3.1 Sample Management and Storage at Clinical Services Program – Leidos Biomedical Research, Inc. (CSP)

Clinical Services Program - Leidos Biomedical Research, Inc.

Attn: Theresa Burks 1050 Boyles Street Bldg. 496/Room 121 Frederick, MD 21702

On days samples are drawn, Jen Bangh at CSP (part of NCI Frederick Central Repositories) should be notified (phone: [301] 846-5893; fax [301] 846-6222). She will arrange same-day courier delivery of the specimens.

All data associated with the participant samples is protected by using a secure database. All Clinical Support Laboratory Staff receive annual training in maintaining records' confidentiality.


All samples drawn at the NIH Clinical Center will be transported to the Clinical Support Laboratory at the Frederick National Laboratory for Cancer Research by couriers.

Samples will be tracked and managed by Central Repository database, where there is no link to personal identifiable information. All samples will be stored in either a -80°C freezer or vapor phase liquid nitrogen. These freezers are located at NCI Frederick Central Repository in Frederick, Maryland.

NCI Frederick Central Repositories (managed under a subcontract) store, among other things, biological specimens in support of NIH clinical studies. All specimens are stored in secure, limited-access facilities with sufficient security, backup, and emergency support capability and monitoring to ensure long-term integrity of the specimens for research.

Specimens are stored in accordance with applicable HHS and FDA Protection of Human Subjects Regulations in accordance with the subcontractor's Federal-wide Assurance. The subcontractor's role limited to clinical research databases and repositories containing participant specimens. The subcontractor does not conduct or have any vested interest in research on human subjects, but does provide services and support the efforts of its customers, many of which are involved in research on human subjects.

It is the intent and purpose of the subcontractor to accept only coded, linked samples and sample information. To the limit of our ability, every effort will be made to ensure that protected information is not sent electronically or by hard copy or on vial labels.

Sample data is stored in the BioSpecimen Inventory System II (BSI). This inventory tracking system is used to manage the storage and retrieval of specimens as well as to maintain specimen data. BSI is designed for controlled, concurrent access. It provides a real-time, multi-user environment for tracking millions of specimens. The system controls how and in what order database updates and searches are performed. This control prevents deadlocks and race conditions. For security, BSI has user password access, 3 types of user access levels, and 36 user permissions (levels of access) that can be set to control access to the system functions. BSI provides audit tracking for processes that are done to specimens including shipping, returning to inventory, aliquoting, thawing, additives, and other processes. BSI tracks the ancestry of specimens as they are aliquoted, as well as discrepancies and discrepancy resolution for specimens received by the repository. If a specimen goes out of the inventory, the system maintains data associated with the withdrawal request. Vials are labeled with a unique BSI ID which is printed in both eye-readable and bar-coded format. No participant -specific information is encoded in this ID.

Investigators are granted view, input, and withdrawal authority only for their specimens. They may not view specimen data or access specimens for which they have not been authorized. Access to specimen storage is confined to repository staff. Visitors to the repositories are escorted by repository staff at all times.

## 5.3.2 Procedures for Storage of Tissue Specimens in the Laboratory of Pathology

Tissues designated for clinical diagnostics are transported to the Laboratory of Pathology (LP) where they are examined grossly and relevant portions are fixed, embedded in paraffin and sectioned and stained for diagnostic interpretation. Unutilized excess tissues are stored for up to three months, in accordance with College of American Pathologists/Joint Commission on Accreditation of Healthcare Organizations (CAP/JCAHO) guidelines, and then discarded.


Following completion of the diagnostic workup, the slides and tissue blocks are stored indefinitely in the LP's clinical archives. All specimens are catalogued and retrieved utilizing the clinical laboratory information systems, in accordance with CAP/JCAHO regulations. The use of any stored specimens for research purposes is only allowed when the appropriate IRB approval has been obtained. In some cases, this approval has been obtained via the original protocol on which the participant was enrolled.

# 5.3.3 Protocol Completion/Sample Destruction

All specimens obtained in the protocol are used as defined in the protocol. Any specimens that are remaining at the completion of the protocol will be stored in the conditions described above. The study will remain open so long as sample or data analysis continues. Samples from consenting subjects will be stored until they are no longer of scientific value or if a subject withdraws consent for their continued use, at which time they will be destroyed. The PI will report any loss or unanticipated destruction of samples per Section 7.2.1. If the patient withdraws consent the participant's data will be excluded from future distributions, but data that have already been distributed for approved research use will not be able to be retrieved.

Samples will also be reported as lost if they are lost in transit between facilities or misplaced by a researcher. Freezer problems, lost samples, or other problems associated with samples that meet expedited reporting requirements (see Section 7.2.1) will also be reported.

#### 6 DATA COLLECTION AND EVALUATION

#### 6.1 DATA COLLECTION

The PI will be responsible for overseeing entry of data into a 21 CFR Part 11-compliant data capture system provided by the NCI CCR and ensuring data accuracy, consistency and timeliness. The principal investigator, associate investigators/research nurses and/or a contracted data manager will assist with the data management efforts. Primary and final analyzed data will have identifiers so that research data can be attributed to an individual human subject participant.

All adverse events, including clinically significant abnormal findings on laboratory evaluations, regardless of severity, will be followed until return to baseline or stabilization of event.

Document AEs from the first study drug administration, Study Day 1 through 28 days after removal from study treatment or until off-study, whichever comes first. Adverse events that are serious need to be recorded through 28 days after the last intervention. Beyond 28 days after the last intervention and through long term follow up (survival of subject), only adverse events which are serious and related to the study intervention need to be recorded.

An abnormal laboratory value will be recorded in the database as an AE **only** if the laboratory abnormality is characterized by any of the following:

- Results in discontinuation from the study
- Is associated with clinical signs or symptoms
- Requires treatment or any other therapeutic intervention
- Is associated with death or another serious adverse event, including hospitalization.
- Is judged by the Investigator to be of significant clinical impact


• If any abnormal laboratory result is considered clinically significant, the investigator will provide details about the action taken with respect to the test drug and about the participant's outcome.

**End of study procedures:** Data will be stored according to HHS, FDA regulations, and NIH Intramural Records Retention Schedule as applicable.

Loss or destruction of data: Should we become aware that a major breach in our plan to protect subject confidentiality and trial data has occurred, this will be reported expeditiously per requirements in Section 7.2.1.

#### **6.2 DATA SHARING PLANS**

# 6.2.1 Human Data Sharing Plan

# What data will be shared?

I will share human data generated in this research for future research as follows:

- Coded, linked data in an NIH-funded or approved public repository.
- Coded, linked data in BTRIS (automatic for activities in the Clinical Center)
- Identified or coded, linked data with approved outside collaborators under appropriate agreements.

#### How and where will the data be shared?

Data will be shared through:

- An NIH-funded or approved public repository: clinicaltrials.gov
- BTRIS (automatic for activities in the Clinical Center).
- Approved outside collaborators under appropriate individual agreements.
- Publication and/or public presentations.

#### When will the data be shared?

- Before publication.
- At the time of publication or shortly thereafter.

# 6.2.2 Genomic Data Sharing Plan

Unlinked genomic data will be deposited in public genomic databases such as dbGaP in compliance with the NIH Genomic Data Sharing Policy.

#### 6.3 RESPONSE CRITERIA

#### 6.3.1 Antitumor Response

Tumor assessments may include the following evaluations: physical examination (with photograph and measurement of skin lesions, as applicable); cross-sectional imaging using computed tomography (CT) or magnetic resonance imaging (MRI) scan of the chest, abdomen, and pelvis (pelvis scan is optional unless known pelvic disease is present at baseline); nuclear bone scan for subjects with known/suspected bone lesions; and CT or MRI scan of the brain (only as clinically warranted based on symptoms/findings). The preferred method of disease assessment is CT with


contrast. If CT with contrast is contraindicated, CT of the chest without contrast and MRI scan of the abdomen/pelvis is preferred.

At baseline, tumor lesions will be selected and categorized as target or non-target lesions. Target lesions include those lesions that can be accurately measured in at least 1 dimension as  $\geq$  20 mm with conventional techniques or  $\geq$  10 mm with CT scan. Malignant lymph nodes with a short axis diameter  $\geq$  15 mm can be considered target lesions. Up to a maximum of 2 target lesions per organ and 5 target lesions in total will be identified at baseline. These lesions should be representative of all involved organs and selected based on their size (those with the longest diameter) and their suitability for accurate repeated measurements. A sum of the longest lesion diameter (LLD) for all target lesions will be calculated and reported as the baseline sum LLD. For malignant lymph nodes identified as target lesions, the short axis diameter will be used in the sum of LLD calculation. All other lesions (or sites of disease) should be identified as non-target lesions (including bone lesions).

All post-baseline response assessments should follow the same lesions identified at baseline. The same mode of assessment (e.g., CT) used to identify/evaluate lesions at baseline should be used throughout the course of the study unless subject safety necessitates a change (e.g., allergic reaction to contrast media).

For the primary endpoint antitumor activity will be evaluated with target and/or non-target lesions according to RECIST Version 1.1.

#### 6.3.2 Disease Parameters

<u>Measurable disease</u>: Measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded) as:

- By chest x-ray:  $\geq$  20 mm;
- By CT scan:
  - O Scan slice thickness 5 mm or under: as > 10 mm
  - Scan slice thickness > 5 mm: double the slice thickness
- With calipers on clinical exam: > 10 mm.

All tumor measurements must be recorded in millimeters (or decimal fractions of centimeters).

Malignant lymph nodes. To be considered pathologically enlarged and measurable, a lymph node must be  $\geq 15$  mm in short axis when assessed by CT scan (CT scan slice thickness recommended to be no greater than 5 mm). At baseline and in follow-up, only the short axis will be measured and followed.

Non-measurable disease. All other lesions (or sites of disease), including small lesions (longest diameter < 10 mm or pathological lymph nodes with  $\ge 10$  to < 15 mm short axis), are considered non-measurable disease. Bone lesions, leptomeningeal disease, ascites, pleural/pericardial effusions, lymphangitis cutis/pulmonitis, inflammatory breast disease, and abdominal masses (not followed by CT or MRI), are considered as non-measurable.


Note: Cystic lesions that meet the criteria for radiographically defined simple cysts should not be considered as malignant lesions (neither measurable nor non-measurable) since they are, by definition, simple cysts.

'Cystic lesions' thought to represent cystic metastases can be considered as measurable lesions, if they meet the definition of measurability described above. However, if non-cystic lesions are present in the same participant, these are preferred for selection as target lesions.

<u>Target lesions</u>. All measurable lesions up to a maximum of 2 lesions per organ and 5 lesions in total, representative of all involved organs, should be identified as **target lesions** and recorded and measured at baseline. Target lesions should be selected on the basis of their size (lesions with the longest diameter), be representative of all involved organs, but in addition should be those that lend themselves to reproducible repeated measurements. It may be the case that, on occasion, the largest lesion does not lend itself to reproducible measurement in which circumstance the next largest lesion which can be measured reproducibly should be selected. A sum of the diameters (longest for non-nodal lesions, short axis for nodal lesions) for all target lesions will be calculated and reported as the baseline sum diameters. If lymph nodes are to be included in the sum, then only the short axis is added into the sum. The baseline sum diameters will be used as reference to further characterize any objective tumor regression in the measurable dimension of the disease.

Non-target lesions. All other lesions (or sites of disease) including any measurable lesions over and above the 5 target lesions should be identified as **non-target lesions** and should also be recorded at baseline. Measurements of these lesions are not required, but the presence, absence, or in rare cases unequivocal progression of each should be noted throughout follow-up.

#### 6.3.3 Methods for Evaluation of Measurable Disease

All measurements should be taken and recorded in metric notation using a ruler or calipers. All baseline evaluations should be performed as closely as possible to the beginning of treatment and never more than 4 weeks before the beginning of the treatment.

The same method of assessment and the same technique should be used to characterize each identified and reported lesion at baseline and during follow-up. Imaging-based evaluation is preferred to evaluation by clinical examination unless the lesion(s) being followed cannot be imaged but are assessable by clinical exam.

<u>Clinical lesions</u>: Clinical lesions will only be considered measurable when they are superficial (e.g., skin nodules and palpable lymph nodes) and  $\geq 10$  mm diameter as assessed using calipers (e.g., skin nodules). In the case of skin lesions, documentation by color photography, including a ruler to estimate the size of the lesion, is recommended.

<u>Chest x-ray</u>: Lesions on chest x-ray are acceptable as measurable lesions when they are clearly defined and surrounded by aerated lung. However, CT is preferable.

<u>Conventional CT and MRI</u>: This guideline has defined measurability of lesions on CT scan based on the assumption that CT slice thickness is 5 mm or less. If CT scans have slice thickness greater than 5 mm, the minimum size for a measurable lesion should be twice the slice thickness. MRI is also acceptable in certain situations (e.g., for body scans).

Use of MRI remains a complex issue. MRI has excellent contrast, spatial, and temporal resolution; however, there are many image acquisition variables involved in MRI, which greatly impact image


quality, lesion conspicuity, and measurement. Furthermore, the availability of MRI is variable globally. As with CT, if an MRI is performed, the technical specifications of the scanning sequences used should be optimized for the evaluation of the type and site of disease. Furthermore, as with CT, the modality used at follow-up should be the same as was used at baseline and the lesions should be measured/assessed on the same pulse sequence. It is beyond the scope of the RECIST guidelines to prescribe specific MRI pulse sequence parameters for all scanners, body parts, and diseases. Ideally, the same type of scanner should be used and the image acquisition protocol should be followed as closely as possible to prior scans. Body scans should be performed with breath-hold scanning techniques, if possible.

# 6.3.4 Response Criteria

All the scans performed at Baseline and other imaging performed as clinically required (other supportive imaging) need to be repeated at subsequent visits. In general, lesions detected at Baseline need to be followed using the same imaging methodology and preferably the same imaging equipment at subsequent tumor evaluation visits.

Brain CT / MRI scan should be performed, if clinically indicated by development of new specific symptoms or on the discretion of the Principal Investigator. For each subject, the Investigator will designate 1 or more of the following measures of tumor status to follow for determining response: CT or MRI images of primary and / or metastatic tumor masses, physical examination findings, and the results of other assessments. All available images collected during the trial period will be considered. The most appropriate measures to evaluate the tumor status of a subject should be used. The measure(s) to be chosen for sequential evaluation during the trial have to correspond to the measures used to document the progressive tumor status that qualifies the subject for enrollment. The tumor response assessment will be assessed and listed according to the Study Calendar 3.5.

The foreseen treatment duration is until disease progression verified by a scan subsequent to the initial documentation of PD, unacceptable toxicity, or any criterion for withdrawal from the trial occurs (see Section 6.3). Before stopping the treatment, progressive disease should be confirmed by imaging 4 to 6 weeks (preferably 6 weeks, but not later) after progression has been diagnosed according to RECIST 1.1 [36]. If progression is based on the occurrence of a new lesion in an area not scanned at Baseline, a further on-study scan 6 weeks later should be considered before performing the 28-Day Safety Follow-up visit. Treatment may be continued despite progression according to RECIST 1.1 at any time if:

- There are no new or concerning symptoms.
- There is no decrease in ECOG PS.
- The Investigator does not consider it necessary to administer a salvage therapy.

The treatment should be stopped immediately, if the subject does not tolerate M7824 or if therapeutic failure occurs, which requires urgent treatment with an additional drug or results in clinically significant progression / deterioration.

Tumor responses to treatment will be assigned based on the evaluation of the response of target, non-target, and new lesions according to RECIST 1.1 (all measurements should be recorded in metric notation).


•To assess objective response, the tumor burden at baseline will be estimated and used for comparison with subsequent measurements. At baseline, tumor lesions will be categorized in target and non-target lesions according to RECIST 1.1.

Results for these evaluations will be recorded with as much specificity as possible so that pre-and post-treatment results will provide the best opportunity for evaluating tumor response.

Any CR or PR should be confirmed according to RECIST 1.1. In the case of a PR or CR, a confirmatory CT or MRI scan should be done no sooner than 4 weeks (preferably at the scheduled 6-week interval).

The Investigator may perform scans in addition to a scheduled trial scan for medical reasons or if the Investigator suspects PD.

As an exploratory endpoint antitumor activity will also be evaluated according to iRECIST [37].

Using iRECIST criteria the following will be incorporated into assessment:

- 1. An increase in the sum of target lesions of more than 20%, unequivocal increase in non-target lesions or new lesions result in iUPD (unconfirmed progressive disease); iUPD can be assigned multiple times as long as iCPD (confirmed progressive disease) is not confirmed at the next assessment.
- 2. Progression is confirmed in the target lesion category if the next imaging assessment after iUPD (4–8 weeks later) confirms a further increase in sum of measures of target disease from iUPD, with an increase of at least 5 mm. Progression is confirmed in the non-target lesion category if subsequent imaging, done 4–8 weeks after iUPD, shows a further unequivocal increase in non-target lesions. Progression is confirmed in the new lesions category if at next assessment additional new lesions appear or an increase in size of previously seen new lesions is seen (≥5 mm for sum of new lesion target).
- 3. However, the criteria for iCPD (after iUPD) are not considered to have been met if complete response, partial response, or stable disease criteria (compared with baseline and as defined by RECIST 1.1) are met at the next assessment after iUPD. The status is reset (unlike RECIST 1.1, in which any progression precludes later complete response, partial response, or stable disease). iCR, iPR, or iSD should then be assigned; and if no change is detected, then the timepoint response is iUPD.
- 6.3.5 Response Criteria by RECIST 1.1

#### 6.3.5.1 Evaluation of Target Lesions

<u>Complete Response (CR)</u>: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.

<u>Partial Response (PR)</u>: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.

<u>Progressive Disease (PD)</u>: At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).


<u>Stable Disease (SD)</u>: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study.

# 6.3.5.2 Evaluation of Non-Target Lesions

<u>Complete Response (CR)</u>: Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).

Note: If tumor markers are initially above the upper normal limit, they must normalize for a participants to be considered in complete clinical response.

Non-CR/Non-PD: Persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits.

<u>Progressive Disease (PD)</u>: Appearance of one or more new lesions and/or *unequivocal progression* of existing non-target lesions. *Unequivocal progression* should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.

Although a clear progression of "non-target" lesions only is exceptional, the opinion of the treating physician should prevail in such circumstances, and the progression status should be confirmed at a later time by the review panel (or Principal Investigator).

# 6.3.5.3 Evaluation of Best Overall Response

The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The participant's best response assignment will depend on the achievement of both measurement and confirmation criteria.

For Participants with Measurable Disease (i.e., Target Disease)

| Target<br>Lesions | Non-Target<br>Lesions | New<br>Lesions | Overall<br>Response | Best Overall Response when Confirmation is Required* |
|---|---|---|---|---|
| CR | CR | No | CR | ≥4 wks. Confirmation** |
| CR | Non-<br>CR/Non-PD | No | PR | |
| CR | Not<br>evaluated | No | PR | ≥4 wks. Confirmation** |
| PR | Non-<br>CR/Non-<br>PD/not<br>evaluated | No | PR | |
| SD | Non-<br>CR/Non-<br>PD/not<br>evaluated | No | SD | Documented at least once ≥4 wks. from baseline** |


| Target<br>Lesions | Non-Target<br>Lesions | New<br>Lesions | Overall<br>Response | Best Overall Response when Confirmation is Required* |
|---|---|---|---|---|
| PD | Any | Yes or<br>No | PD | |
| Any | PD*** | Yes or<br>No | PD | no prior SD, PR or CR |
| Any | Any | Yes | PD | |

- \* See RECIST 1.1 manuscript for further details on what is evidence of a new lesion.
- \*\* Only for non-randomized trials with response as primary endpoint.
- \*\*\* In exceptional circumstances, unequivocal progression in non-target lesions may be accepted as disease progression.

Note: Participants with a global deterioration of health status requiring discontinuation of treatment without objective evidence of disease progression at that time should be reported as "symptomatic deterioration." Every effort should be made to document the objective progression even after discontinuation of treatment.

# For Participants with Non-Measurable Disease (i.e., Non-Target Disease)

| Non-Target Lesions | New Lesions | Overall Response |
|--------------------|-------------|------------------|
| CR | No | CR |
| Non-CR/non-PD | No | Non-CR/non-PD* |
| Not all evaluated | No | not evaluated |
| Unequivocal PD | Yes or No | PD |
| Any | Yes | PD |

<sup>\* &#</sup>x27;Non-CR/non-PD' is preferred over 'stable disease' for non-target disease since SD is increasingly used as an endpoint for assessment of efficacy in some trials so to assign this category when no lesions can be measured is not advised

### 6.3.5.4 Duration of Response

<u>Duration of overall response</u>: The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).


The duration of overall CR is measured from the time measurement criteria are first met for CR until the first date that progressive disease is objectively documented.

<u>Duration of stable disease</u>: Stable disease is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started, including the baseline measurements.

# 6.3.5.5 Progression-Free Survival

PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.

#### 6.4 TOXICITY CRITERIA

The following adverse event management guidelines are intended to ensure the safety of each participants while on the study. The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for AE reporting. All appropriate treatment areas should have access to a copy of the CTCAE version 5.0. A copy of the CTCAE version 5.0 can be downloaded from the CTEP web site (http://ctep.cancer.gov/protocolDevelopment/electronic applications/ctc.htm).

# 7 NIH REPORTING REQUIREMENTS / DATA AND SAFETY MONITORING PLAN

#### 7.1 **DEFINITIONS**

Please refer to definitions provided in Policy 801: Reporting Research Events found at: <a href="https://irbo.nih.gov/confluence/pages/viewpage.action?pageId=36241835#Policies&Guidance-800Series-ComplianceandResearchEventReportingRequirements">https://irbo.nih.gov/confluence/pages/viewpage.action?pageId=36241835#Policies&Guidance-800Series-ComplianceandResearchEventReportingRequirements</a>.

# 7.2 OHSRP OFFICE OF COMPLIANCE AND TRAINING / IRB REPORTING

# 7.2.1 Expedited Reporting

Please refer to the reporting requirements in Policy 801: Reporting Research Events and Policy 802 Non-Compliance Human Subjects Research found at: <a href="https://irbo.nih.gov/confluence/pages/viewpage.action?pageId=36241835#Policies&Guidance-800Series-ComplianceandResearchEventReportingRequirements">https://irbo.nih.gov/confluence/pages/viewpage.action?pageId=36241835#Policies&Guidance-800Series-ComplianceandResearchEventReportingRequirements</a>.

Note: Only IND Safety Reports that meet the definition of an unanticipated problem will need to be reported per these policies.

# 7.2.2 IRB Requirements for PI Reporting at Continuing Review

Please refer to the reporting requirements in Policy 801: Reporting Research Events found at: <a href="https://irbo.nih.gov/confluence/pages/viewpage.action?pageId=36241835#Policies&Guidance-800Series-ComplianceandResearchEventReportingRequirements">https://irbo.nih.gov/confluence/pages/viewpage.action?pageId=36241835#Policies&Guidance-800Series-ComplianceandResearchEventReportingRequirements</a>.

#### 7.2.3 NCI Clinical Director Reporting

Problems expeditiously reviewed by the OHSRP in the NIH eIRB system will also be reported to the NCI Clinical Director/designee; therefore, a separate submission for these reports is not necessary.


In addition to those reports, all deaths that occur within 30 days after receiving a research intervention should be reported via email unless they are due to progressive disease.

To report these deaths, please send an email describing the circumstances of the death to <a href="https://www.ncircumstances.ncircumstances">NCICCRQA@mail.nih.gov</a> within one business day of learning of the death.

# 7.3 NIH REQUIRED DATA AND SAFETY MONITORING PLAN

## 7.3.1 Principal Investigator/Research Team

The clinical research team will meet on a regular basis (approximately weekly) when participants are being actively treated on the trial to discuss each participant. Decisions about dose level enrollment and dose escalation if applicable will be made based on the toxicity data from prior participants.

All data will be collected in a timely manner and reviewed by the principal investigator or a lead associate investigator. Events meeting requirements for expedited reporting as described in Section 7.2.2 will be submitted within the appropriate timeline.

The principal investigator will review adverse event and response data on each participant to ensure safety and data accuracy. The principal investigator will personally conduct or supervise the investigation and provide appropriate delegation of responsibilities to other members of the research staff.

# 7.3.2 Data Safety Monitoring Board (DSMB) (OSRO)

The DSMB is an independent group of at least 3 experts that monitors participant safety and advises The Sponsor. DSMB members will be separate and independent of study staff participating in this trial and should not have scientific, financial, or other conflicts of interest related to this trial. The DSMB will consist of members with appropriate expertise to contribute to the interpretation of data from this trial. A quorum will consist of a simple majority.

The DSMB will review cumulative safety data from this trial at least annually.

The DSMB will meet as requested by the sponsor or PI.

The DSMB will have a final review meeting at the end of the study.

Procedures for DSMB reviews/meetings will be defined in the DSMB charter. The DSMB will review applicable data, including, but not limited to, enrollment, demographics, dosing data, clinical laboratory data, and safety data, at scheduled timepoints during this trial as defined in the DSMB charter. The DSMB will review blinded aggregate data in the open session of the DSMB meetings.

Additional data may be requested by the DSMB, and interim statistical reports may be generated as deemed necessary and appropriate by the Sponsor. As an outcome of each review/meeting, the DSMB will make a recommendation as to the advisability of proceeding with study product administration, and to continue, modify, or terminate this trial.


#### 8 SPONSOR PROTOCOL/SAFETY REPORTING

#### 8.1 **DEFINITIONS**

#### 8.1.1 Adverse Event

Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event (AE) can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product (ICH E6 (R2)).

#### 8.1.2 Adverse Event of Special Interest (AESI)

Mucosal bleeding events which are at least possibly related to study drug (M7824) will be captured as AESIs. These events will not require expedited reporting to the study sponsor unless they also meet SAE criteria.

## 8.1.3 Serious Adverse Event (SAE)

An adverse event or suspected adverse reaction is considered serious if in the view of the investigator or the sponsor, it results in any of the following:

- Death:
- A life-threatening adverse event (see Section 8.1.4);
- Inpatient hospitalization or prolongation of existing hospitalization
  - O A hospitalization/admission that is pre-planned (i.e., elective or scheduled surgery arranged prior to the start of the study), a planned hospitalization for pre-existing condition, or a procedure required by the protocol, without a serious deterioration in health, is not considered a serious adverse event.
  - A hospitalization/admission that is solely driven by non-medical reasons (e.g., hospitalization for patient convenience) is not considered a serious adverse event.
  - o Emergency room visits or stays in observation units that do not result in admission to the hospital would not be considered a serious adverse event. The reason for seeking medical care should be evaluated for meeting one of the other serious criteria.
- Persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions;
- A congenital anomaly/birth defect;
- Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered a serious adverse drug experience when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.


### 8.1.4 Life-threatening

An adverse event or suspected adverse reaction is considered "life-threatening" if, in the view of either the investigator or sponsor, its occurrence places the patient or subject at immediate risk of death. It does not include an adverse event or suspected adverse reaction that, had it occurred in a more severe form, might have caused death (21CFR312.32).

# 8.1.5 Severity

The severity of each Adverse Event will be assessed utilizing the CTCAE version 5.0.

# 8.1.6 Relationship to Study Product

All AEs will have their relationship to study product assessed using the terms: related or not related.

- Related There is a reasonable possibility that the study product caused the adverse event. Reasonable possibility means that there is evidence to suggest a causal relationship between the study product and the adverse event.
- <u>Not Related</u> There is not a reasonable possibility that the administration of the study product caused the event.

# 8.1.7 Adverse Events of Special Interest (AESI)

An adverse event of special interest (AESI) is one of scientific and medical interest specific to understanding of the Investigational Product(s) and may require close monitoring and rapid communication by the investigator to the sponsor. An AESI may be serious or non-serious. The rapid reporting of AESIs allows ongoing surveillance of these events to characterize and understand them in association with the use of these investigational products.

Only AESIs that match the definition of SAE will be reported as other SAEs within 24 hours from the knowledge of event.

The following adverse events, regardless of site, will be collected as an AESI to enable evaluation of potential risk factors, such as site/past radiation/associated infection at site/recent instrumentation and other variables such as time to onset, exposure history, grade of bleeding, anatomical sites, etc. can be collected.

# 8.2 ASSESSMENT OF SAFETY EVENTS

AE information collected will include event description, date of onset, assessment of severity and relationship to study product and alternate etiology (if not related to study product), date of resolution of the event, seriousness and outcome. The assessment of severity and relationship to the study product will be done only by those with the training and authority to make a diagnosis and listed on the Form FDA 1572 as the site principal investigator or sub-investigator. AEs occurring during the collection and reporting period will be documented appropriately regardless of relationship. AEs will be followed through resolution.

SAEs will be:


• Assessed for severity and relationship to study product and alternate etiology (if not related to study product) by a licensed study physician listed on the Form FDA 1572 as the site principal investigator or sub-investigator.

- Recorded on the appropriate SAE report form, the medical record and captured in the clinical database.
- Followed through resolution by a licensed study physician listed on the Form FDA 1572 as the site principal investigator or sub-investigator.

For timeframe of recording adverse events, please refer to Section 6.1. All serious adverse events recorded must be reported to the sponsor. All serious adverse events recorded from the time of first investigational product administration must be reported to the sponsor with the exception of any listed in section 8.4.

#### 8.3 REPORTING OF SERIOUS ADVERSE EVENTS

Any AE that meets protocol-defined serious criteria or meets the definition of Adverse Event of Special Interest that require expedited reporting must be submitted immediately (within 24 hours of awareness) to OSRO Safety using the CCR SAE report form. Any exceptions to the expedited reporting requirements are found in section **8.4**.

All SAE reporting must include the elements described in Section 8.2.

SAE reports will be submitted to the Center for Cancer Research (CCR) at: OSROSafety@mail.nih.gov and to the CCR PI and study coordinator. CCR SAE report form and instructions can be found at: https://ccrod.cancer.gov/confluence/display/CCRCRO/Forms+and+Instructions

Following the assessment of the SAE by OSRO, other supporting documentation of the event may be requested by the OSRO Safety and should be provided as soon as possible.

#### 8.4 WAIVER OF EXPEDITED REPORTING TO CCR

As overall survival, which includes death due to disease progression and hospitalization due to disease progression are part of the study objectives, and captured as an endpoint in this study, death/hospitalization due to disease progression will not be reported in expedited manner to the sponsor. However, if there is evidence suggesting a causal relationship between the study drug and the event, report the event in an expedited manner according to Section **8.3**.

#### 8.5 SAFETY REPORTING CRITERIA TO THE PHARMACEUTICAL COLLABORATORS

Reporting will be per the collaborative agreement.

#### 8.6 REPORTING PREGNANCY

All required pregnancy reports/follow-up to OSRO will be submitted to: <u>OSROSafety@mail.nih.gov</u> and to the CCR PI and study coordinator. Forms and instructions can be found here: https://ccrod.cancer.gov/confluence/display/CCRCRO/Forms+and+Instructions

# 8.6.1 Maternal exposure

If a participant becomes pregnant during the course of the study, the study treatment should be discontinued immediately, and the pregnancy reported to the Sponsor. The potential risk of exposure of the fetus to the investigational agent(s) or chemotherapy agents (s) should be documented in box B5 of the MedWatch form "Describe Event or Problem".

Pregnancy itself is not regarded as an SAE. However, congenital abnormalities or birth defects and spontaneous miscarriages that meet serious criteria (Section 8.1.3) should be reported as SAEs.

The outcome of all pregnancies should be followed up and documented.

# 8.6.2 Paternal exposure

Male participants should refrain from fathering a child or donating sperm during the study and for 2 months after the last dose of M7824.

Pregnancy of the participant's partner is not considered to be an AE. The outcome of all pregnancies occurring from the date of the first dose until 2 months after the last dose should, if possible, be followed up and documented. Pregnant partners may be offered the opportunity to participate in an institutional pregnancy registry protocol (e.g., the NIH IRP pregnancy registry study) to provide data about the outcome of the pregnancy for safety reporting purposes.

## 8.7 REGULATORY REPORTING FOR STUDIES CONDUCTED UNDER CCR-SPONSORED IND

Following notification from the investigator, CCR, the IND sponsor, will report any suspected adverse reaction that is both serious and unexpected in expedited manner to the FDA in accordance to 21 CFR 31.2.32. CCR will report an AE as a suspected adverse reaction only if there is evidence to suggest a causal relationship between the study product and the adverse event. CCR will notify FDA and all participating investigators (i.e., all investigators to whom the sponsor is providing drug under its INDs or under any investigator's IND) in an IND safety report of potential serious risks from clinical trials or any other source, as soon as possible, in accordance to 21 CFR Part 312.32.

All serious events will be reported to the FDA at least annually in a summary format.

## 8.8 SPONSOR PROTOCOL DEVIATION REPORTING

A Protocol Deviation is defined as any non-compliance with the clinical trial Protocol, Manual of Operational Procedures (MOP) and other Sponsor approved study related documents, GCP, or protocol-specific procedural requirements on the part of the participant, the Investigator, or the study site staff inclusive of site personnel performing procedures or providing services in support of the clinical trial.

It is the responsibility of the study Staff to document any protocol deviation identified by the Staff or the site Monitor in the CCR Protocol Deviation Tracking System (PDTS) online application. The entries into the PDTS online application should be timely, complete, and maintained per CCR PDTS user requirements.

In addition, any deviation to the protocol should be documented in the participant's source records and reported to the reviewing IRB per their guidelines. OSRO required protocol deviation


reporting is consistent with E6(R2) GCP: Integrated Addendum to ICH E6(R1): 4.5 Compliance with Protocol; 5.18.3 (a), and 5.20 Noncompliance; and ICH E3 16.2.2 Protocol deviations.

# 9 CLINICAL MONITORING PLAN

Clinical site monitoring is conducted to ensure:

- that the rights of the participants are protected;
- that the study is implemented per the approved protocol, Good Clinical Practice and standard operating procedures; and,
- the quality and integrity of study data and data collection methods are maintained.

Monitoring for this study will be performed by NCI CCR Office of Sponsor and Regulatory Oversight (OSRO) Sponsor and Regulatory Oversight Support (SROS) Services contractor. Clinical site monitoring activities will be based on OSRO standards, FDA Guidance E6(R2) Good Clinical Practice: Integrated Addendum to ICH E6(R1) March 2018, and applicable regulatory requirements.

Details of clinical site monitoring will be documented in a Clinical Monitoring Plan (CMP) developed by OSRO. CMPs will be protocol-specific, risk-based and tailored to address human subject protections and integrity of the study data. OSRO will determine the intensity and frequency of monitoring based on several factors, including study type, phase, risk, complexity, expected enrollment rate, and any unique attributes of the study and the site. The Sponsor will conduct a periodic review of the CMP to confirm the plan's continued appropriateness. A change to the protocol, significant or pervasive non-compliance with GCP, or the protocol may trigger CMP updates.

OSRO SROS Monitoring visits and related activities will be conducted throughout the life cycle of each protocol. The first activity is before the study starts to conduct a Site Assessment Visit (SAV) (as warranted), followed by a Site Initiation Visit (SIV), Interim Monitoring Visit(s) (IMVs), and a study Close-Out Visit (COV).

Some monitoring activities may be performed remotely, while others will occur at the study site. Monitoring visit reports will describe visit activities, observations, and associated action items or follow-up required for resolution of any issues, discrepancies, or deviations. Monitoring reports will be distributed to the study PI, NCI CCR QA, CCR Protocol Support Office, coordinating center (if applicable), and the OSRO regulatory file.

The site Monitor will inform the study team of any deviations observed during monitoring visits. If unresolved, the Monitor will request that the site Staff enter the deviations in the CCR Protocol Deviation Tracking System (PDTS) for deviation reporting to the Sponsor and as applicable per institutional and IRB guidance.

## 10 STATISTICAL CONSIDERATIONS

#### 10.1 STATISTICAL HYPOTHESIS

The primary objective of this trial is to determine the objective response rate of combination immunotherapy in participants with HPV associated malignancies. A secondary hypothesis (objective) will be to obtain preliminary data on duration of response, PFS, OS and ratio of


participants that are hospitalized because of adverse events attributed to disease progression. An exploratory hypothesis (objective) will be to evaluate exploratory immunologic studies to understand and improve the administered treatment.

In patients with cervical cancer with prior pelvic radiation and boost brachytherapy, a key secondary objective is to evaluate the safety of the combination at a reduced dose level in these patients where a potential higher risk of grade 3 hematuria may exist with the full starting doses of M7824 at 1200 mg and NHS-IL12 at 16.8 mcg/kg.

## 10.2 SAMPLE SIZE DETERMINATION

Data from the ongoing trial indicates that a response rate for M7824 may be approximately 30%. In the main study cohort (Cohort 1), this trial will try to demonstrate if the proposed combination therapies may be associated with an improved response rate.

The trial will treat participants with HPV related cancers with HPV vaccine + M7824 + NHS-IL12. The objective is to determine if this treatment can be associated with an acceptable response rate. To establish the efficacy of this combination treatment, the primary objective would be to determine if using the proposed agents would rule out a 30% response rate and result in a response rate consistent with 60%. As such, this trial in participants with HPV associated malignancies will be conducted using a Simon optimal two-stage phase II trial design (Simon R, Controlled Clinical Trials 10:1-10, 1989) to rule out an unacceptably low PR+CR rate of 30% (p0=0.30) in favor of an improved response rate of 60% (p1=0.60). With alpha=0.10 (probability of accepting a poor treatment=0.10) and beta = 0.10 (probability of rejecting a good treatment=0.10), the first stage will enroll 8 evaluable checkpoint naïve participants, and if 0 to 2 of the 8 have a clinical response, then no further participants will be accrued. If 3 or more of the first 8 checkpoint naïve participants have a response, then accrual would continue until a total of 20 evaluable checkpoint naïve participants have been treated. As it may take up to several months to determine if a patient has experienced a response, a temporary pause in the accrual may be necessary to ensure that enrollment to the second stage is warranted. If there are 3 to 8 checkpoint naïve participants with a response out of 20 participants, this would be an uninterestingly low response rate. If there were 9 or more of 20 (45.0%) checkpoint naïve patients who experienced a response, this would be sufficiently interesting to warrant possible further study of the combination in later trials in this disease type; decisions about future use of the combination will incorporate response as well as toxicity profile information. Under the null hypothesis (30% response rate), the probability of early termination is 55.2%.

In the cohort with patients with cervical cancer with prior pelvic radiation and boost brachytherapy where a potential higher risk of grade 3 hematuria may exist with the full starting doses of M7824 at 1200 mg and NHS-IL12 at 16.8 mcg/kg, the safety evaluation may require up to 12 patients as outlined in Section 3.4.3, and if there are preliminary hints of efficacy within these 12 patients, up to 12 additional patients may be enrolled at the dose found to be safe for these patients to further explore the safety as well as the potential response rate in a small number of patients.

It is expected that if 2 participants per month enroll on the trial, in order to enroll up to a total of 20 evaluable participants with checkpoint naïve disease in the main cohort, and 12+12=24 maximum in the patients in cohort 2, up to 3 years may be required. To allow for several inevaluable participants for the primary objective and potential replacements based on HPV status the accrual ceiling will be set at 56 participants. If additional patients are required to enroll on the


trial to account for screen failures and inevaluable patients, the ceiling increase will be incorporated in an amendment.

#### 10.3 POPULATIONS FOR ANALYSES

All participants who receive any investigational treatment will be evaluable for safety and toxicity evaluations. All participants will be evaluable for toxicity from the time of their first treatment with any agent.

For efficacy, a modified intention to treat population will be used. Only those participants who have measurable disease present at baseline and have had their disease re-evaluated will be considered evaluable for response. (Note: Participants who exhibit objective disease progression prior to the end of cycle 1 will also be considered evaluable.)

### 10.4 STATISTICAL ANALYSES

# 10.4.1 General Approach

Participants will be evaluated with respect to the grades and types of toxicities obtained. The results will be presented descriptively and tabled if appropriate. Further planned analyses are described below.

# 10.4.2 Analysis of the Primary Endpoints

The percentage of checkpoint naïve subjects whose initial doses of study drugs are not modified that achieve an objective confirmed complete or partial overall tumor response using RECIST Version 1.1 will be evaluated. If anti-tumor responses are observed, the 95% confidence interval of the response rate will be evaluated.

## 10.4.3 Analysis of the Secondary Endpoints

Data will be obtained on duration of response, PFS, OS and ratio of participants that are hospitalized because of adverse events attributed to disease progression. In addition, patients in cohort 2 will have their safety evaluated based on the description in Section 3.4.3.

# 10.4.3.1 Duration of Response

The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that PD is objectively documented and is evaluated using the Kaplan-Meier method.

#### 10.4.3.2 Progression-Free Survival

PFS will be evaluated using Kaplan-Meier methods. PFS will be defined as the time from the date of first treatment to the date of disease progression or death (any cause) whichever occurs first. Subjects who do not have disease progression or have not died at the end of follow up will be censored at the last known date the subject was progression free.

# 10.4.3.3 Objective Response

Objective response is a complete or partial radiographic response as defined by RECIST 1.1 (Section 6.3.5).


## 10.4.3.4 Overall Survival

OS will be evaluated using Kaplan-Meier methods. OS will be defined as the time from the date of first treatment to the date of death (any cause). Subjects who are alive at the end of follow up will be censored at the last known date alive.

# 10.4.4 Safety Analyses

Safety endpoints will be analyzed as summary statistics during treatment and/or as change scores from baseline assessments. AEs will be coded as defined in the Medical Dictionary for Regulatory Activities (MedDRA). All AEs will be recorded and tabulated following each treatment. AEs will be recorded by severity, frequency, and relationship to the study intervention and will be presented by System Organ Class (SOC) designations and preferred term groupings. Information on each AE will include start date, stop date, severity, relationship, expectedness, outcome, and duration. Adverse events leading to premature discontinuation from the study intervention and serious treatment-emergent AEs will be presented either in a Table or a Listing.

In addition, overall safety will be assessed by descriptive analyses using tabulated frequencies of AEs by grade using CTCAE Version 5 within dose cohorts and for the overall study population in terms of treatment-emergent AEs, SAEs, and clinically significant changes in safety laboratory tests, physical examinations, ECGs, and vital signs.

Patients in cohort 2 will have their safety evaluated as detailed in Section 3.4.3, with up to 12 patients, with further evaluation focusing on bleeding events in the maximum of 12 patients enrolled at the dose considered safe among the patients in this cohort also being enrolled for an exploratory evaluation of efficacy.

# 10.4.5 Baseline Descriptive Statistics

Baseline Characteristics will be described.

## 10.4.6 Planned Interim Analyses

Interim assessment of efficacy will be made according to the Simon two stage phase II designs of each cohort described in Section 10.4.6.

## 10.4.7 Tabulation of Individual Participant Data

Individual responses in a cohort may be depicted within a larger group using a waterfall plot or spider diagram.

# 10.4.8 Exploratory Analyses

## 10.4.8.1 Exploratory Analyses: Immune Responses

Where feasible exploratory immune analyses will be conducted to evaluate anti-tumor immune responses. Immune response will be assessed among all subjects treated in each cohort. The magnitude of immune responses will be described. A subject will be considered evaluable for immune response if they receive at least one dose of treatment. The percentage of subjects with a positive immune response will be evaluated by cohort. For flow cytometry analyses on PBMC samples, Student T tests or Kruskal-Wallis and Wilcoxon rank sum tests as appropriate will be performed on percentages of TNF- $\alpha$  and/or IFN- $\gamma$  expressing cells among the different cohorts to determine any significant differences in cell populations. For antigen specific T cell responses, a positive immune response is defined by CMI reactivity in *ex vivo* stimulation using a flow


cytometric readout (cytokine production or CD107 expression). Antigen-specific peptide challenge assays require a readout of >250 reactive T-cells/million cells above the background [38].

10.4.8.2 Exploratory Analyses: Preliminary Activity in Patients Receiving Lower Doses

In patients who receive reduced initial doses of therapy as per Section 3.4.3, both in the dose seeking portion as well as in a small group of patients treated at the safe dose, the percentage of subjects who achieve an objective confirmed complete or partial overall tumor response using RECIST Version 1.1 for a specific initial dose will be evaluated. If anti-tumor responses are observed, the 95% confidence interval of the response rate will be evaluated.

## 11 COLLABORATIVE AGREEMENTS

# 11.1 COOPERATIVE RESEARCH AND DEVELOPMENT AGREEMENT (CRADA)

A CRADA (02666) is in place with EMD Serono for the supply of M7824 and NHS-IL12.

A CRADA (03279) is in place with PDS Biotechnology for the supply of PDS0101.

### 12 HUMAN SUBJECTS PROTECTIONS

## 12.1 RATIONALE FOR SUBJECT SELECTION

Subjects from all racial/ethnic groups are eligible for this study if they meet the eligibility criteria. Efforts will be made to extend accrual to a representative population. Due to impaired cellular immunity which may affect the efficacy of treatment, patients with poorly controlled HIV as well as patents with detectable viral loads of hepatitis B and C will be excluded.

Participants who do not accept blood transfusions will be excluded. As there is a risk of severe bleeding with this study drug, participants must be willing to receive blood transfusions if medically necessary for their own safety.

#### 12.2 Participation of Children

Individuals under the age of 18 will not be eligible to participate in this study because of unknown toxicities in pediatric patients.

## 12.3 PARTICIPATION OF SUBJECTS UNABLE TO GIVE CONSENT

Adults unable to provide consent are excluded from enrolling in the protocol. However, it is possible that subjects enrolled in the protocol may permanently lose the capacity to consent for themselves during the course of this study. In the event this occurs, the subjects will remain in the study because there is a prospect of direct benefit from research participation. All subjects ≥ age 18 will be offered the opportunity to fill in their wishes for research and care, and assign a substitute decision maker on the "NIH Advance Directive for Health Care and Medical Research Participation" form so that another person can make decisions about their medical care in the event that they become incapacitated or cognitively impaired during the course of the study.

Note: The PI or AI will contact the NIH Ability to Consent Assessment Team (ACAT) for evaluation to assess ongoing capacity of the subjects and to identify an LAR, as needed.


Please see Section 12.5.1 for consent procedure.

#### 12.4 RISKS/BENEFIT ASSESSMENT

Participants will receive evaluation of their disease at the National Cancer Institute's Clinical Center. The potential benefit to a participant that goes onto study is a reduction in the bulk of their tumor which may or may not have a favorable impact on symptoms and/or survival.

Potential adverse reactions attributable to the administration of the study drug utilized in this trial are discussed in Section 14. All care will be taken to minimize side effects, but they can be unpredictable in nature and severity. Participants will be examined and evaluated prior to enrollment. All evaluations to monitor the treatment of participants will be recorded in the medical record. If participants suffer any physical injury as a result of the participation in this study, immediate medical treatment is available at the Clinical Center, National Cancer Institute, Bethesda, Maryland.

Although no compensation is available, any injury will be evaluated and treated in keeping with the benefits or care to which participants are entitled under applicable regulations.

#### 12.4.1 Risks

Some of the procedures performed on this study are not known to be associated with risk. These include urine tests and EKGs. Below are a list of procedures and study interventions that are associated with risk.

# 12.4.1.1 Study Drug Risks

Risks include the possible occurrence of any of a range of side effects which are listed in the Consent Document.

Participants may be harmed from being in this study by toxicity due to the drug or combination of drugs given during this study. M7824 is similar to immune check point inhibitors. There are preliminary data to suggest that not all patients benefit from immune check point inhibitors nor M7824. Additionally, there are preliminary data to suggest that an unexpectedly rapid progression of disease occurs in some patients receiving immunotherapy such as immune checkpoint inhibitors.

## 12.4.1.2 Risk of Optional Biopsies

All care will be taken to minimize risks that may be incurred by tumor sampling. However, there are procedure-related risks (such as bleeding, infection and visceral injury) that will be explained fully during informed consent.

# 12.4.1.3 Risks of Exposure to Ionizing Radiation

This research study involves the possibility of 7 CT CAP scans, 1 brain CT scan, and 2 CT guided biopsies collected for research purposes.

The amount of radiation exposure you will receive from these procedures is equal to approximately 9.4 rem. The CT scans and CT guided biopsies in this study will expose the research participant to 31.3 years' worth of background radiation. This level of exposure results in an increased risk of cancer.


#### 12.4.1.4 Additional Risks of CT Scans

In addition to the radiation risks addressed above, CT scans that employ contrast may cause allergic reactions, injection site reactions abdominal discomfort and fainting.

#### 12.4.1.5 Research Blood Collection Risks

Risks of blood draws include pain and bruising in the area where the needle is placed, lightheadedness, and rarely, fainting. When large amounts of blood are collected, low red blood cell count (anemia) can develop.

#### 12.4.1.6 Other Risks

Risks include the possible occurrence of any of a range of side effects which are listed in the Consent Document or this protocol document. Frequent monitoring for adverse effects will help to minimize the risks associated with administration of the study agents.

### 12.4.2 Benefits

The potential benefit to a patient that goes onto study is a reduction in the bulk of their tumor which may or may not have favorable impact on symptoms and/or survival.

## 12.4.3 Assessment of Potential Risks and Benefits

Metastatic or refractory/recurrent HPV associated malignancies (cervical, anal, oropharyngeal cancers, etc.) are in need of improved therapy options. Preclinical studies suggest that the use of a combination of multiple immunotherapy agents may have improved anti-tumor efficacy.

A number of clinically appropriate strategies to minimize risks to participants have been built into the protocol through the means of inclusion/exclusion criteria, monitoring strategies, and management guidelines. Overall, there is direct potential benefit of the combination of a therapeutic vaccine against HPV positive cancers (PDS0101), a tumor targeted immunocytokine (NHS-IL12) and a bifunctional fusion protein targeting PD-L1 and TGF beta (M7824) in subjects with advanced HPV associated malignancies for participants retaining the ability to consent and those who lose capacity to consent during the course of the trial with this combination immunotherapy proposed in this study.

The potential benefit to a participant that goes onto this study is a reduction in the bulk of their tumor which may or may not have favorable impact on symptoms and/or survival.

Potential adverse reactions attributable to the administration of the study drug utilized in this trial are discussed in Section 14. All care will be taken to minimize side effects, but they can be unpredictable in nature and severity.

#### 12.5 CONSENT PROCESS AND DOCUMENTATION

The informed consent document will be provided as a physical or electronic document to the participant or consent designee(s) as applicable for review prior to consenting. A designated study investigator will carefully explain the procedures and tests involved in this study, and the associated risks, discomforts and benefits. In order to minimize potential coercion, as much time as is needed to review the document will be given, including an opportunity to discuss it with friends, family members and/or other advisors, and to ask questions of any designated study investigator. A signed informed consent document will be obtained prior to entry onto the study.


The initial consent process as well as re-consent, when required, may take place in person or remotely (e.g., via telephone or other NIH approved remote platforms used in compliance with policy, including HRPP Policy 303) per discretion of the designated study investigator and with the agreement of the participant/consent designee(s). Whether in person or remote, the privacy of the subject will be maintained. Consenting investigators (and participant/consent designee, when in person) will be located in a private area (e.g., clinic consult room). When consent is conducted remotely, the participant/consent designee will be informed of the private nature of the discussion and will be encouraged to relocate to a more private setting if needed.

Consent will be documented with required signatures on the physical document (which includes the printout of an electronic document sent to participant) or as described below, with a manual (non-electronic) signature on the electronic document. When required, witness signature will be obtained similarly as described for the investigator and participant.

# Manual (non-electronic) signature on electronic document:

When a manual signature on an electronic document is used for the documentation of consent at the NIH Clinical Center, this study will use the following to obtain the required signatures:

- Adobe platform (which is not 21 CFR Part 11 compliant); or,
- iMedConsent platform (which is 21 CFR Part 11 compliant)

During the consent process, participants and investigators will view individual copies of the approved consent document on screens at their respective locations (if remote consent); the same screen may be used when at the same location, but is not required.

Both the investigator and the subject will sign the document using a finger, stylus or mouse.

Note: Refer to the CCR SOP PM-2, Obtaining and Documenting the Informed Consent Process for additional information (e.g., verification of participant identity when obtaining consent remotely) found at <a href="https://ccrod.cancer.gov/confluence/pages/viewpage.action?pageId=73203825">https://ccrod.cancer.gov/confluence/pages/viewpage.action?pageId=73203825</a>.

As there is an optional biopsy for research in this protocol, the participant will be asked to sign a separate consent at the time of the procedure. If the participant refuses the optional biopsy at that time, the refusal will be documented in the medical record and in the research record.

# 12.5.1 Consent Process for Participants Who Decline Other Treatment Options

Participants who are eligible because they decline the treatment options described in the eligibility criteria (see Section 2.1) will have consent obtained in the presence of an independent consent monitor from the Bioethics department or Human Subjects Protection Unit (HSPU).

12.5.2 Consent Process for Adults Who Lack Capacity to Consent to Research Participation

For participants addressed in Section 12.3, an LAR will be identified consistent with Policy 403 and informed consent obtained from the LAR, as described in Section 12.5.


## 13 REGULATORY AND OPERATIONAL CONSIDERATIONS

#### 13.1 STUDY DISCONTINUATION AND CLOSURE

This study may be temporarily suspended or prematurely terminated if there is sufficient reasonable cause. Written notification, documenting the reason for study suspension or termination, will be provided by the suspending or terminating party to study participants, investigator, the Investigational New Drug (IND) and regulatory authorities. If the study is prematurely terminated or suspended, the Principal Investigator (PI) will promptly inform study participants, the Institutional Review Board (IRB), and sponsor and will provide the reason(s) for the termination or suspension. Study participants will be contacted, as applicable, and be informed of changes to study visit schedule.

Circumstances that may warrant termination or suspension include, but are not limited to:

- Determination of unexpected, significant, or unacceptable risk to participants
- Demonstration of efficacy that would warrant stopping
- Insufficient compliance to protocol requirements
- Data that are not sufficiently complete and/or evaluable
- Determination that the primary endpoint has been met
- Determination of futility

Study may resume once concerns about safety, protocol compliance, and data quality are addressed, and satisfy the sponsor, IRB and as applicable, Food and Drug Administration (FDA).

# 13.2 QUALITY ASSURANCE AND QUALITY CONTROL

Each clinical site will perform internal quality management of study conduct, data and biological specimen collection, documentation and completion. An individualized quality management plan will be developed to describe a site's quality management.

Quality control (QC) procedures will be implemented beginning with the data entry system and data QC checks that will be run on the database will be generated. Any missing data or data anomalies will be communicated to the site(s) for clarification/resolution.

Following written Standard Operating Procedures (SOPs), the monitors will verify that the clinical trial is conducted, and data are generated and biological specimens are collected, documented (recorded), and reported in compliance with the protocol, International Conference on Harmonisation Good Clinical Practice (ICH GCP), and applicable regulatory requirements (e.g., Good Laboratory Practices (GLP), Good Manufacturing Practices (GMP)).

The investigational site will provide direct access to all trial related sites, source data/documents, and reports for the purpose of monitoring and auditing by the sponsor, and inspection by local and regulatory authorities.

#### 13.3 CONFLICT OF INTEREST POLICY

The independence of this study from any actual or perceived influence, such as by the pharmaceutical industry, is critical. Therefore, any actual conflict of interest of persons who have a role in the design, conduct, analysis, publication, or any aspect of this trial will be disclosed and managed. Furthermore, persons who have a perceived conflict of interest will be required to have such conflicts managed in a way that is appropriate to their participation in the design and conduct


of this trial. The study leadership in conjunction with the National Cancer Institute has established policies and procedures for all study group members to disclose all conflicts of interest and will establish a mechanism for the management of all reported dualities of interest.

## 13.4 CONFIDENTIALITY AND PRIVACY

Participant confidentiality and privacy is strictly held in trust by the participating investigators, their staff, and the sponsor(s). This confidentiality is extended to cover testing of biological samples and genetic tests in addition to the clinical information relating to participants. Therefore, the study protocol, documentation, data, and all other information generated will be held in strict confidence. No information concerning the study or the data will be released to any unauthorized third party without prior written approval of the sponsor.

All research activities will be conducted in as private a setting as possible.

The study monitor, other authorized representatives of the sponsor, representatives of the Institutional Review Board (IRB), and/or regulatory agencies may inspect all documents and records required to be maintained by the investigator, including but not limited to, medical records (office, clinic, or hospital) and pharmacy records for the participants in this study. The clinical study site will permit access to such records.

The study participant's contact information will be securely stored at the clinical site for internal use during the study. At the end of the study, all records will continue to be kept in a secure location for as long a period as dictated by the reviewing IRB, Institutional policies, or sponsor requirements.

Study participant research data, which is for purposes of statistical analysis and scientific reporting, will be stored at the NCI CCR. This will not include the participant's contact or identifying information. Rather, individual participants and their research data will be identified by a unique study identification number. The study data entry and study management systems used by the clinical site and by NCI CCR research staff will be secured and password protected. At the end of the study, all study databases will be archived at the NIH.

To further protect the privacy of study participants, a Certificate of Confidentiality has been issued by the National Institutes of Health (NIH). This certificate protects identifiable research information from forced disclosure. It allows the investigator and others who have access to research records to refuse to disclose identifying information on research participation in any civil, criminal, administrative, legislative, or other proceeding, whether at the federal, state, or local level. By protecting researchers and institutions from being compelled to disclose information that would identify research participants, Certificates of Confidentiality help achieve the research objectives and promote participation in studies by helping assure confidentiality and privacy to participants.

### 14 PHARMACEUTICAL INFORMATION

## 14.1 PDS0101 (IND # 019267)

14.1.1 Source / Acquisition and Accountability

PDS0101 will be provided by PDS Biotechnology through a CRADA.


R-DOTAP and HPVmix will be provided to the clinical trial site by the manufacturer. The investigator or designee (e.g., pharmacist) will maintain an ongoing inventory of the investigational product supply according to standard site procedures. The investigational product will be dispensed at the direction of an investigator for administration to a study participant enrolled on the clinical trial. Disposal of expired or unused product will be returned to the manufacturer or disposed of according to standard site procedures based on agreement between the manufacturer and the site.

# 14.1.2 Toxicity

In 2014-2016, a Phase I/IIA human clinical trial was performed at 3 sites in the US in 12 subjects with high-risk HPV infection and biopsy-proven CIN1 to study the safety and immunogenicity of PDS0101. Administration of PDS0101 was well tolerated. The majority of AEs were due to administration site reactions. Most administration site reactions were mild or moderate in severity. Some more severe administration site reactions including swelling and redness were reported in the 3- and 10-mg R-DOTAP cohorts. Most administration site reactions resolved the same day or within a few days. Per the subject symptom diary, administration site reactions were more severe and of longer duration in subjects in the 10-mg R-DOTAP cohort. No clinically significant differences in the types and pattern of TEAEs were observed between Vaccinations 1, 2, or 3. No DLTs were observed; thus, the MTD was the 10-mg R-DOTAP dose. No serious adverse events (SAEs), study discontinuations due to adverse events, or deaths occurred. No clinically relevant abnormal hematology, blood chemistry, urinalysis, or physical findings were observed.

# 14.1.3 Formulation and Preparation

PDS0101 is a 2-vial formulation which is mixed 1:1 v/v just prior to administration.

<u>Vial #1 (ImmunoMAPK-RDOTAP)</u>: is a sterile, turbid pharmaceutical suspension of liposomal nanoparticles composed of the pure R-enantiomer of the cationic (positively charged) lipid DOTAP (dioleoyl-trimethylammonium propane). The particle size is between 100-200nm. RDOTAP is a novel immune modulator which induces the production of important cytokines and chemokines and also enhances the cytolytic T-Lymphocyte response when combined with the antigenic peptides. ImmunoMAPK-RDOTAP is has been evaluated at 3 dose levels, 1.0, 3.0 and 10.0mg.

<u>Vial #2 (HPVmix)</u>: is a sterile, clear and slightly viscous suspension consisting of 6 nononcogenic lipidated peptides selected from immunogenic regions of the human papillomavirus strain 16 E6 and E7 proteins. The peptides exist in a mixed micellar particulate state. The HPVmix formulation contains 20% by volume of dimethyl sulfoxide (DMSO). HPVmix is being evaluated at a single dose level of 2.7 mg.

The 1:1 mixture of R-DOTAP and HPVmix (antigens) yields a mixture of liposomes and peptide mixed micelles in 10% DMSO. The nanoparticulate vaccine induces antigen specific T-cell therapeutic responses.

# 14.1.4 Stability and Storage

# ImmunoMAPK-RDOTAP (Vial #1) and HPV Mix (Vial #2)

Storage: Store at  $-70^{\circ}$ C  $\pm 10^{\circ}$ C.


Shipping: Shipped on dry ice in insulated container. Always check the

temperature monitoring device to ensure maintenance of required

storage condition during shipment.

R-DOTAP Thawing: Place at room temperature for a minimum of 90 minutes (1.5 hours)

prior to mixing with HPVmix.

HPVmix Thawing: Remove from freezer at least 60 minutes (1 hour) after removal of

RDOTAP. Place at room temperature for a minimum of 30 minutes (0.5 hours) and a maximum of 90 minutes (1.5 hours) prior to mixing

with RDOTAP.

Mixture: PDS0101 should not be administered if held in vial for more than

120 minutes (2 hours) at ambient temperature after mixing.

### 14.1.5 Administration Procedures

Subcutaneous administration in a limb. Each subsequent vaccination should preferably be administered alternating between limbs (e.g., L arm  $\rightarrow$  R arm).

Two separate 0.5mL injections preferably ~ 6 cm apart of vaccine in the same extremity

Total Dose: 3.0mg R-DOTAP/2.7 mg HPV Peptides

# 14.1.6 Incompatibilities

Not available.

# 14.2 M7824 (MSB0011359C) (IND # 019267)

## 14.2.1 Source / Acquisition and Accountability

M7824 is manufactured and supplied for the trial by EMD Serono Research and Development Institute.

M7824 will be provided to the clinical trial site by the manufacturer. The investigator or designee (e.g., pharmacist) will maintain an ongoing inventory of the investigational product supply according to standard site procedures. The investigational product will be dispensed at the direction of an investigator for administration to a study participant enrolled on the clinical trial. Disposal of expired or unused product will be returned to the manufacturer or disposed of according to standard site procedures based on agreement between the manufacturer and the site.

# 14.2.2 Toxicity

The immunoglobulin portion of M7824 molecule is identical to avelumab (Bavencio). Respective warnings and precautions for grade 2 or higher immune-mediated pneumonitis, immune-mediated colitis, immune-mediated endocrinopathies, immune-mediated hepatitis) and infusion reactions are included in the prescribing for Bavencio (bavencio.com). Participants will be pre-medicated to prophylax against infusions reactions. The following additionally significant immune-mediated adverse reactions have occurred in less than 1% of 1738 participants treated with BAVENCIO: myocarditis with fatal cases, myositis, psoriasis, arthritis, exfoliative dermatitis, erythema multiforme, pemphigoid, hypopituitarism, uveitis, Guillain-Barré syndrome, and systemic


inflammatory response. The above irAEs are all considered an anticipated risk of treatment with M7824 and thus will not be considered DLTs.

In a phase 1, open-label 3+3 dose-escalation study of M7824 in 16 participants, 3 participants experienced grade 3 drug-related adverse events including skin infection secondary to grade 2 bullous pemphigoid, lipase increased, and colitis with associated anemia. There were no grade 4 – 5 treatment related adverse events. Please see table below for details.


# **Treatment-related adverse events**

| | 3 mg/kg (n = 3) | | 10 mg/kg (n=3) | | 20 mg/kg (n=7) | | $Total\ (n=16)$ | |
|---|---|---|---|---|---|---|---|---|
| | Any | Grade | Any | Grade | Any | Grade | Any | Grade |
| D 4' ' 4 '41 | Grade | 3 | Grade | 3 | Grade | 3 | Grade | 3 |
| Participants with any event** | 2<br>(66.7) | (33.3) | (33.3) | 0 (0.0) | 4<br>(57.1) | 2<br>(28.6) | 7<br>(43.8) | 3<br>(18.8) |
| Anemia | (00.7) | (33.3) | (33.3) | | 1 (14.3) | 1 (14.3) | 1 (6.3) | 1 (6.3) |
| Bullous pemphigoid | 1 (33.3) | | | | | | 1 (6.3) | |
| Colitis | | | | | 1 (14.3) | 1 (14.3) | 1 (6.3) | 1 (6.3) |
| Dermatitis acneiform | | | 1 (33.3) | | | | 1 (6.3) | |
| Dyspnea exertional*** | | | | | 1 (14.3) | | 1 (6.3) | |
| Hyperthyroidism | | | | | 1 (14.3) | | 1 (6.3) | |
| Hypophosphatemia | | | | | 1 (14.3) | | 1 (6.3) | |
| Hypothyroidism | | | (33.3) | | 1<br>(14.3) | | 2<br>(12.5) | |
| Infusion-related reaction | | | | | 1<br>(14.3) | | 1 (6.3) | |
| Keratoacanthoma | | | | | 1<br>(14.3) | | 1 (6.3) | |
| Lipase increase | | | | | 1 (14.3) | 1 (14.3) | 1 (6.3) | 1 (6.3) |
| Nausea | 1 (33.3) | | | | | | 1 (6.3) | |
| Pruritus | 1 (33.3) | | | | | | 1 (6.3) | |
| Rash maculo-<br>papular | 1 (33.3) | | 1 (33.3) | | | | 2<br>(12.5) | |
| Skin infection | 1 (33.3) | 1 (33.3) | | | | | 1 (6.3) | 1 (6.3) |
| Vomiting | (33.3) | | | | | | 1 (6.3) | |

<sup>\*\*</sup>There were no treatment-related AEs in the 3 participants treated with 1 mg/kg M7824.

<sup>\*\*\*</sup>The differential for this dyspnea was pneumonitis vs. lymphangitic spread of disease (disease progression).


As of August 2017, > 500 participants have been treated with M7824 across multiple solid tumor expansion cohorts. The safety profile is consistent with other monotherapy checkpoint inhibitors, with the exception of keratoacanthomas and cutaneous squamous cell carcinomas which have occurred in approximately 3-5% of participants and are well managed with surgical excision. These lesions have not been a criterion for treatment discontinuation, but thus far have all spontaneously regressed following treatment discontinuation.



At least 2 instances of nodular regenerative hyperplasia have been observed with the use of this agent.

# 14.2.2.1 Hemophagocytic lymphohistiocytosis (HLH)

HLH/MAS is an inflammatory response which may be related to immune therapy, but the mechanism is poorly understood. This may present with liver function test abnormalities, low blood cell counts, fevers, elevated ferritin and/or elevated triglycerides. HLH may be acquired (secondary), but in the setting of immune therapy we believe it is acquired. This can spontaneously resolve or be treated with steroids or other immune suppressive therapies.

## 14.2.3 Formulation and Preparation

M7824 is provided as a sterile liquid formulation and packaged at a 10 mg/mL concentration in USP/ Ph Eur type I 50R vials that are filled with drug product solution to allow an extractable volume of 60 mL (600 mg/60 mL). The vials are closed with rubber stoppers in serum format complying with USP and Ph Eur with an aluminum crimp seal closure. Each single-use vial contains 600mg of M7824, formulated as 10mg/mL of active, 6% (w/v) Trehalose, 40 mM NaCl, 5 mM Methionine, 0.05% (w/v) Tween 20, 10 mM L-Histidine at pH 5.5.

The liquid formulation is diluted directly with 0.9% sodium chloride solution for injection. The estimated volumes of delivery are anticipated to be no more than 250mL. The verified concentration range in the infusion solution is 0.16 mg/mL to 9.6 mg/mL.

### 14.2.4 Stability and Storage

M7824 must be stored at 2°C to 8°C until use. Product stored at room temperature for extended periods of time might be subject to degradation. M7824 must not be frozen. Rough shaking of the reconstituted solution must be avoided.

The chemical and physical in-use stability for the infusion solution of M7824 in 0.9% sodium chloride for injection has been demonstrated for a total of 72 hours at room temperature; however, from a microbiological point of view, the diluted solution should be used immediately and is not


intended to be stored unless dilution has taken place in controlled and validated aseptic conditions. No other drugs should be added to the infusion containers containing M7824. See Manual of Preparation of approved ancillary supplies.

## 14.2.5 Administration Procedures

See Section 3.2.

14.2.6 Incompatibilities

Not available.

# 14.3 NHS-IL12 (IND # 019267)

# 14.3.1 Source / Acquisition and Accountability

NHS-IL12 is manufactured and supplied by EMD Serono.

NHS-IL12 will be provided to the clinical trial site by the manufacturer. The investigator or designee (e.g., pharmacist) will maintain an ongoing inventory of the investigational product supply according to standard site procedures. The investigational product will be dispensed at the direction of an investigator for administration to a study participant enrolled on the clinical trial. Disposal of expired or unused product will be returned to the manufacturer or disposed of according to standard site procedures based on agreement between the manufacturer and the site.

# 14.3.2 Toxicity

Subjects (n=59) were treated subcutaneously with NHS-IL12 in a single ascending dose cohort followed by a multiple ascending dose cohort (n=37 with every 4-week dosing). The primary objective of this trial was to determine MTD as defined by the number of DLTs. None of the subjects treated with single or multiple doses up to 12.0 µg/kg experienced a DLT. At 16.8 µg/kg, 1/6 subjects had a DLT (grade 3 increase in alanine transaminase [ALT]). At 21.8 μg/kg, 2/6 subjects had a DLT (grade 3 increase in aspartate transaminase [AST] and ALT; grade 3 increase in lipase without clinical signs of pancreatitis). MTD was 16.8 µg/kg. The most frequently observed treatment-related adverse event (TRAE) was decreased lymphocyte count (27/59 subjects; 45.8%). Other TRAEs included decreased white blood cells (WBCs) (24/59; 40.7%), fever and elevated AST (21 each; 35.6%), elevated ALT (20; 3.9%), and anemia and flu-like symptoms (18 each; 30.5%) (Table 2; Supplemental Figure 5). Among the cohort receiving 16.8 μg/kg, the most frequently reported TRAEs were elevated AST (75%), decreased WBCs and elevated ALT (68.8% each), and decreased lymphocyte count and fever (62.5% each). At least one grade  $\geq$  3 TRAE was seen in 12/59 subjects (20.3%). These included decreased lymphocyte count (5; 8.5%), decreased neutrophil count (4; 6.8%), elevated ALT (3; 5.1%), decreased WBCs (2; 3.4%), and hypokalemia, hyperhidrosis, elevated alkaline phosphatase, AST, and lipase (1 each; 1.7%). All grade  $\geq$  3 TRAEs were transient; only hyperhidrosis was symptomatic. One grade 4 TRAE was observed (asymptomatic decreased lymphocyte count); no grade 5 TRAE was observed.

## 14.3.3 Formulation and Preparation

NHS-IL12 is formulated as a 1.5 mg/mL solution and is supplied by the Sponsor in single-use glass vials with a rubber stopper and sealed with an aluminum Flip Off® crimp seal closure.


The contents of the NHS-IL12 vials are sterile and nonpyrogenic, and do not contain bacteriostatic preservatives. Any spills that occur should be cleaned up using the facility's standard cleanup procedures for biologic products.

Rough shaking of the solution must be avoided.

NHS-IL12 drug product will be administered undiluted (1500mcg/mL) for doses  $\geq$  300mcg. However, for doses below 300 µg, NHS-IL12 drug product must be diluted with 0.9% saline solution (sodium chloride injection). Doses 100 to 299 mcg will be administered as a 500mcg/mL solution and doses 30 to 99 mcg will be administered as a 150 mcg/mL solution. Detailed information on medical devices to be used for the preparation and administration of NHS-IL12 will be provided in the Investigator Brochure.

Any unused portion of the solution should be discarded in biohazard waste disposal with final disposal by accepted local and national standards of incineration.

# 14.3.4 Stability and Storage

NHS-IL12 drug product must be stored at 2°C to 8°C until use, with a temperature log maintained daily. All medication boxes supplied to the study site must be stored carefully, safely, and separately from other drugs.

The chemical and physical in-use stability of NHS-IL12 diluted and undiluted solution in syringes has been demonstrated for 24 hours at 25°C. However, to reduce the risk of microbial contamination, the solution should be used immediately unless medication preparation has been performed in controlled and validated aseptic conditions. Rough shaking of the solution must be avoided.

#### 14.3.5 Administration Procedures

NHS-IL12 is administered subcutaneously. It can be given in the arm, leg or abdomen. Where feasible it should be given in a different limb than the vaccine.

## 14.3.6 Incompatibilities

Not available.


#### 15 REFERENCES

- 1. Viens LJ, Henley SJ, Watson M, Markowitz LE, Thomas CC, Thompson TD, Razzaghi H, Saraiya M: **Human Papillomavirus-Associated Cancers United States, 2008-2012**. *MMWR Morb Mortal Wkly Rep* 2016, **65**(26):661-666.
- 2. Long HJ, 3rd, Bundy BN, Grendys EC, Jr., Benda JA, McMeekin DS, Sorosky J, Miller DS, Eaton LA, Fiorica JV, Gynecologic Oncology Group S: Randomized phase III trial of cisplatin with or without topotecan in carcinoma of the uterine cervix: a Gynecologic Oncology Group Study. *J Clin Oncol* 2005, 23(21):4626-4633.
- 3. Vermorken JB, Mesia R, Rivera F, Remenar E, Kawecki A, Rottey S, Erfan J, Zabolotnyy D, Kienzer HR, Cupissol D *et al*: **Platinum-based chemotherapy plus cetuximab in head and neck cancer**. *N Engl J Med* 2008, **359**(11):1116-1127.
- 4. Long HJ, 3rd: **Management of metastatic cervical cancer: review of the literature**. *J Clin Oncol* 2007, **25**(20):2966-2974.
- 5. Eng C, Chang GJ, You YN, Das P, Rodriguez-Bigas M, Xing Y, Vauthey JN, Rogers JE, Ohinata A, Pathak P *et al*: **The role of systemic chemotherapy and multidisciplinary management in improving the overall survival of patients with metastatic squamous cell carcinoma of the anal canal**. *Oncotarget* 2014, **5**(22):11133-11142.
- 6. Monk BJ, Sill MW, McMeekin DS, Cohn DE, Ramondetta LM, Boardman CH, Benda J, Cella D: Phase III trial of four cisplatin-containing doublet combinations in stage IVB, recurrent, or persistent cervical carcinoma: a Gynecologic Oncology Group study. *J Clin Oncol* 2009, 27(28):4649-4655.
- 7. Tewari KS, Sill MW, Long HJ, 3rd, Penson RT, Huang H, Ramondetta LM, Landrum LM, Oaknin A, Reid TJ, Leitao MM *et al*: **Improved survival with bevacizumab in advanced cervical cancer**. *N Engl J Med* 2014, **370**(8):734-743.
- 8. Monk BJ, Sill MW, Burger RA, Gray HJ, Buekers TE, Roman LD: **Phase II trial of bevacizumab in the treatment of persistent or recurrent squamous cell carcinoma of the cervix: a gynecologic oncology group study.** *J Clin Oncol* 2009, **27**(7):1069-1074.
- 9. van Herpen CM, van der Voort R, van der Laak JA, Klasen IS, de Graaf AO, van Kempen LC, de Vries IJ, Boer TD, Dolstra H, Torensma R *et al*: Intratumoral rhIL-12 administration in head and neck squamous cell carcinoma patients induces B cell activation. *Int J Cancer* 2008, 123(10):2354-2361.
- 10. Grohmann U, Belladonna ML, Bianchi R, Orabona C, Ayroldi E, Fioretti MC, Puccetti P: IL-12 acts directly on DC to promote nuclear localization of NF-kappaB and primes DC for IL-12 production. *Immunity* 1998, 9(3):315-323.
- 11. Del Vecchio M, Bajetta E, Canova S, Lotze MT, Wesa A, Parmiani G, Anichini A: Interleukin-12: biological properties and clinical application. *Clin Cancer Res* 2007, 13(16):4677-4685.
- 12. Massarelli E, William W, Johnson F, Kies M, Ferrarotto R, Guo M, Feng L, Lee JJ, Tran H, Kim YU *et al*: **Combining Immune Checkpoint Blockade and Tumor-Specific**


Vaccine for Patients With Incurable Human Papillomavirus 16-Related Cancer: A Phase 2 Clinical Trial. *JAMA Oncol* 2019, **5**(1):67-73.

- 13. Lonez C, Vandenbranden M, Ruysschaert JM: Cationic liposomal lipids: from gene carriers to cell signaling. *Prog Lipid Res* 2008, 47(5):340-347.
- 14. Wood L, et al.: In: Society for Immunotherapy of Cancer (SITC): November 8, 2019 2019; National Harbor, MD.
- 15. Boyerinas B, Jochems C, Fantini M, Heery CR, Gulley JL, Tsang KY, Schlom J: Antibody-Dependent Cellular Cytotoxicity Activity of a Novel Anti-PD-L1 Antibody Avelumab (MSB0010718C) on Human Tumor Cells. Cancer Immunol Res 2015, 3(10):1148-1157.
- 16. Heery CR, O'Sullivan-Coyne G, Madan RA, Cordes L, Rajan A, Rauckhorst M, Lamping E, Oyelakin I, Marte JL, Lepone LM *et al*: **Avelumab for metastatic or locally advanced previously treated solid tumours (JAVELIN Solid Tumor): a phase 1a, multicohort, dose-escalation trial**. *Lancet Oncol* 2017, **18**(5):587-598.
- 17. Donahue RN, Lepone LM, Grenga I, Jochems C, Fantini M, Madan RA, Heery CR, Gulley JL, Schlom J: **Analyses of the peripheral immunome following multiple administrations of avelumab, a human IgG1 anti-PD-L1 monoclonal antibody**. *J Immunother Cancer* 2017, 5:20.
- 18. Blobe GC, Schiemann WP, Lodish HF: **Role of transforming growth factor beta in human disease**. *N Engl J Med* 2000, **342**(18):1350-1358.
- 19. Dumont N, Arteaga CL: **Transforming growth factor-beta and breast cancer: Tumor promoting effects of transforming growth factor-beta**. *Breast Cancer Res* 2000, **2**(2):125-132.
- 20. Formenti SC, Lee P, Adams S, Goldberg JD, Li X, Xie MW, Ratikan JA, Felix C, Hwang L, Faull KF *et al*: Focal Irradiation and Systemic TGFbeta Blockade in Metastatic Breast Cancer. *Clin Cancer Res* 2018, **24**(11):2493-2504.
- 21. Ivanovic V, Melman A, Davis-Joseph B, Valcic M, Geliebter J: **Elevated plasma levels** of TGF-beta 1 in patients with invasive prostate cancer. *Nat Med* 1995, 1(4):282-284.
- 22. Shen M, Tsai Y, Zhu R, Keng PC, Chen Y, Chen Y, Lee SO: **FASN-TGF-beta1-PD-L1** axis contributes to the development of resistance to NK cell cytotoxicity of cisplatin-resistant lung cancer cells. *Biochim Biophys Acta Mol Cell Biol Lipids* 2018, 1863(3):313-322.
- 23. Tsushima H, Kawata S, Tamura S, Ito N, Shirai Y, Kiso S, Imai Y, Shimomukai H, Nomura Y, Matsuda Y *et al*: **High levels of transforming growth factor beta 1 in patients with colorectal cancer: association with disease progression**. *Gastroenterology* 1996, **110**(2):375-382.
- 24. Terabe M, Robertson FC, Clark K, De Ravin E, Bloom A, Venzon DJ, Kato S, Mirza A, Berzofsky JA: Blockade of only TGF-beta 1 and 2 is sufficient to enhance the efficacy of vaccine and PD-1 checkpoint blockade immunotherapy. *Oncoimmunology* 2017, 6(5):e1308616.


25. Vanpouille-Box C, Formenti SC: **Dual Transforming Growth Factor-beta and Programmed Death-1 Blockade: A Strategy for Immune-Excluded Tumors?** *Trends Immunol* 2018, **39**(6):435-437.

- 26. Grenga I, Donahue RN, Gargulak ML, Lepone LM, Roselli M, Bilusic M, Schlom J: Anti-PD-L1/TGFbetaR2 (M7824) fusion protein induces immunogenic modulation of human urothelial carcinoma cell lines, rendering them more susceptible to immune-mediated recognition and lysis. *Urol Oncol* 2018, 36(3):93 e91-93 e11.
- 27. Jochems C, Tritsch SR, Pellom ST, Su Z, Soon-Shiong P, Wong HC, Gulley JL, Schlom J: **Analyses of functions of an anti-PD-L1/TGFbetaR2 bispecific fusion protein** (M7824). *Oncotarget* 2017, 8(43):75217-75231.
- 28. Knudson KM, Hicks KC, Luo X, Chen JQ, Schlom J, Gameiro SR: M7824, a novel bifunctional anti-PD-L1/TGFbeta Trap fusion protein, promotes anti-tumor efficacy as monotherapy and in combination with vaccine. *Oncoimmunology* 2018, 7(5):e1426519.
- 29. Lan Y, Zhang D, Xu C, Hance KW, Marelli B, Qi J, Yu H, Qin G, Sircar A, Hernandez VM et al: Enhanced preclinical antitumor activity of M7824, a bifunctional fusion protein simultaneously targeting PD-L1 and TGF-beta. Sci Transl Med 2018, 10(424).
- 30. Ravi R, Noonan KA, Pham V, Bedi R, Zhavoronkov A, Ozerov IV, Makarev E, A VA, Wysocki PT, Mehra R *et al*: **Bifunctional immune checkpoint-targeted antibody-ligand traps that simultaneously disable TGFbeta enhance the efficacy of cancer immunotherapy**. *Nat Commun* 2018, **9**(1):741.
- 31. David JM, Dominguez C, McCampbell KK, Gulley JL, Schlom J, Palena C: A novel bifunctional anti-PD-L1/TGF-beta Trap fusion protein (M7824) efficiently reverts mesenchymalization of human lung cancer cells. *Oncoimmunology* 2017, 6(10):e1349589.
- 32. Strauss J, Heery C, Schlom J, Madan RA, Cao L, Kang Z, Lamping E, Marte JL, Donahue RN, Grenga I et al: Phase 1 trial of M7824 (MSB0011359C), a bifunctional fusion protein targeting PD-L1 and TGF-beta, in advanced solid tumors. Clin Cancer Res 2018.
- 33. Fallon J, Tighe R, Kradjian G, Guzman W, Bernhardt A, Neuteboom B, Lan Y, Sabzevari H, Schlom J, Greiner JW: **The immunocytokine NHS-IL12 as a potential cancer therapeutic**. *Oncotarget* 2014, **5**(7):1869-1884.
- 34. Strauss J, Heery CR, Kim JW, Jochems C, Donahue RN, Montgomery AS, McMahon S, Lamping E, Marte JL, Madan RA *et al*: **First-in-Human Phase I Trial of a Tumor-Targeted Cytokine (NHS-IL12) in Subjects with Metastatic Solid Tumors**. *Clin Cancer Res* 2019, **25**(1):99-109.
- 35. Lepone LM, Donahue RN, Grenga I, Metenou S, Richards J, Heery CR, Madan RA, Gulley JL, Schlom J: Analyses of 123 Peripheral Human Immune Cell Subsets:

  Defining Differences with Age and between Healthy Donors and Cancer Patients
  Not Detected in Analysis of Standard Immune Cell Types. *J Circ Biomark* 2016, 5:5.


36. Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M *et al*: **New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1)**. *Eur J Cancer* 2009, **45**(2):228-247.

- 37. Seymour L, Bogaerts J, Perrone A, Ford R, Schwartz LH, Mandrekar S, Lin NU, Litiere S, Dancey J, Chen A *et al*: **iRECIST: guidelines for response criteria for use in trials testing immunotherapeutics**. *Lancet Oncol* 2017, **18**(3):e143-e152.
- 38. Zhestianikov VD, Savel'eva GE, Kalinin VL: [The adaptive response to mitomycin C exposure in the hyper-radioresistant mutant Escherichia coli Gamr444].

Adaptivnyi otvet na vozdeistvie mitomitsinom C u giperradiorezistentnogo mutanta Escherichia coli Gamr444. *Tsitologiia* 1991, **33**(1):88-96.


# 16 APPENDICIES

# 16.1 APPENDIX A PERFORMANCE STATUS CRITERIA

| ECOG Performance Status Scale | | Karnofsky Performance Scale | |
|---|---|---|---|
| Grade | Descriptions | Percent | Description |
| 0 | Normal activity. Fully active, | 100 | Normal, no complaints, no evidence of disease. |
| | able to carry on all pre-disease performance without restriction. | 90 | Able to carry on normal activity; minor signs or symptoms of disease. |
| 1 | Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able | 80 | Normal activity with effort; some signs or symptoms of disease. |
| | to carry out work of a light or<br>sedentary nature (e.g., light<br>housework, office work). | 70 | Cares for self, unable to carry on normal activity or to do active work. |
| 2 | In bed <50% of the time. Ambulatory and capable of all self-care, but unable to carry out | 60 | Requires occasional assistance, but is able to care for most of his/her needs. |
| | any work activities. Up and about more than 50% of waking hours. | 50 | Requires considerable assistance and frequent medical care. |
| 3 | In bed >50% of the time. Capable of only limited self-care, | 40 | Disabled, requires special care and assistance. |
| | confined to bed or chair more than 50% of waking hours. | 30 | Severely disabled, hospitalization indicated. Death not imminent. |
| 4 | 100% bedridden. Completely disabled. Cannot carry on any | 20 | Very sick, hospitalization indicated. Death not imminent. |
| | self-care. Totally confined to bed or chair. | 10 | Moribund, fatal processes progressing rapidly. |
| 5 | Dead. | 0 | Dead. |